## Johnson & Johnson Vision Care, Inc.

# Clinical Study Protocol

# Characterizing Successful Myopic Multifocal Contact Lens Wearers

Protocol CR-5945

Version: 9.0 Amendment 8

Date: 20 December 2019

Investigational Products: etafilcon A Daily Disposable Multifocal Contact Lens

Key Words: Daily Disposable Multifocal contact lens, successful lens wear, habitual contact lens, soft contact lens, distance vision, intermediate vision, near vision, contact lens drop out

#### Statement of Compliance to protocol, GCP and applicable regulatory guidelines:

This trial will be conducted in compliance with the protocol, ISO 14155,<sup>1</sup> the International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP),<sup>2</sup> the Declaration of Helsinki,<sup>3</sup> and all applicable regulatory requirements.

#### **Confidentiality Statement:**

This document contains confidential information, which should not be copied, referred to, released or published without written approval from Johnson & Johnson Vision Care. The information may not be disclosed to others except to the extent necessary to obtain Institutional Review Board/Independent Ethics Committee approval and informed consent, or as required by International, Federal and State Laws, as applicable. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed without the written permission of Johnson & Johnson Vision Care. Any supplemental information that may be added to this document is also confidential and proprietary to Johnson & Johnson Vision Care and must be kept in confidence in the same manner as the contents of this document.

#### **TABLE OF CONTENTS**

| PROTO | COL TITLE, NUMBER, VERSION | 7 |
|---|---|---|
| SPONS | OR NAME AND ADDRESS | 7 |
| MEDIC | AL MONITOR | 7 |
| AUTHO | DRIZED SIGNATURES | 8 |
| CHANG | GE HISTORY | 10 |
| SYNOP | PSIS | 13 |
| COMM | ONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS | 24 |
| 1. IN | TRODUCTION AND BACKGROUND | 26 |
| 1.1. | Name and Descriptions of Investigational Products | 26 |
| 1.2. | Intended Use of Investigational Products | 26 |
| 1.3. | Summary of Findings from Nonclinical Studies | 26 |
| 1.4. | Summary of Known Risks and Benefits to Human Subjects | 26 |
| 1.5.<br>Clinic | Relevant Literature References and Prior Clinical Data Relevant to Proposed cal Study | 26 |
| | UDY OBJECTIVES, ENDPOINTS AND HYPOTHESES | |
| 2.1. | Objectives | |
| 2.2. | Endpoints | |
| 2.3. | Hypotheses | |
| 3. TA | ARGETED STUDY POPULATION | |
| 3.1. | General Characteristics | 28 |
| 3.2. | Inclusion Criteria | 28 |
| 3.3. | Exclusion Criteria | 29 |
| 3.4. | Enrollment Strategy | 30 |
| 4. ST | UDY DESIGN AND RATIONALE | 30 |
| 4.1. | Description of Study Design | 30 |
| 4.2. | Study Design Rationale | 30 |
| 4.3. | Enrollment Target and Study Duration | 31 |
| 5. TE | ST ARTICLE ALLOCATION AND MASKING | 31 |
| 5.1. | Test Article Allocation | 31 |
| 5.2. | Masking | 31 |
| 5.3. | Procedures for Maintaining and Breaking the Masking | 31 |
| 6. ST | UDY INTERVENTION | 32 |
| 6.1. | Identity of Test Articles. | 32 |
| 6.2 | Ancillary Supplies/Products | 32 |

| 6.3. Administration of Test Articles | 32 |
|--------------------------------------------------------------------|------|
| 6.4. Packaging and Labeling | 33 |
| 6.5. Storage Conditions | |
| 6.6. Collection and Storage of Samples | 33 |
| 6.7. Accountability of Test Articles | 33 |
| 7. STUDY EVALUATIONS | 34 |
| 7.1. Time and Event Schedule | 34 |
| 7.1.1. Additional screening visits | 34 |
| 7.2. Detailed Study Procedures | 34 |
| VISIT 1 39 | |
| VISIT 2 42 | |
| VISIT 3 47 | |
| VISIT 4 51 | |
| VISIT 5 55 | |
| VISIT 6 58 | |
| Final Evaluation | 60 |
| 7.3. Unscheduled Visits | 61 |
| 7.4. Laboratory Procedures | 64 |
| 8. SUBJECTS COMPLETION/WITHDRAWAL | |
| 8.1. Completion Criteria | 64 |
| 8.2. Withdrawal/Discontinuation from the Study | 64 |
| 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION | 65 |
| 10. DEVIATIONS FROM THE PROTOCOL | 66 |
| 11. STUDY TERMINATION | 66 |
| 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS | 66 |
| 13. ADVERSE EVENTS | 68 |
| 13.1. Definitions and Classifications | 68 |
| 13.2. Assessing Adverse Events | 70 |
| 13.2.1. Causality Assessment | 70 |
| 13.2.2. Severity Assessment | 70 |
| 13.3. Documentation and Follow-Up of Adverse Events | 71 |
| 13.4. Reporting Adverse Events | 72 |
| 13.4.1. Reporting Adverse Events to Sponsor | 72 |
| 13.4.2. Reporting Adverse Events to the Responsible IEC/IRB and He | alth |


| 13.4.3. Event of Special Interest | 73 |
|---|---|
| 13.5. Reporting of Pregnancy | 73 |
| 14. STATISTICAL METHODS | 74 |
| 14.1. General Considerations | 74 |
| 14.2. Sample Size Justification | 74 |
| 14.3. Analysis Populations | 74 |
| 14.4. Level of Statistical Significance. | 75 |
| 14.5. Primary Analysis | 75 |
| 14.6. Secondary Analysis | 75 |
| 14.7. Other Exploratory Analyses | 75 |
| 14.8. Interim Analysis | 75 |
| 14.9. Procedure for Handling Missing Data and Drop-Outs | 75 |
| 14.10. Procedure for Reporting Deviations from Statistical Plan | 76 |
| 15. DATA HANDLING AND RECORD KEEPING/ARCHIVING | 76 |
| 15.1. Electronic Case Report Form/Data Collection | 76 |
| 15.2. Subject Record | 77 |
| 16. DATA MANAGEMENT | 77 |
| 16.1. Access to Source Data/Document | 77 |
| 16.2. Confidentiality of Information | 77 |
| 16.3. Data Quality Assurance | 78 |
| 17. MONITORING | 78 |
| 18. ETHICAL AND REGULATORY ASPECTS | 78 |
| 18.1. Study-Specific Design Considerations | 78 |
| 18.2. Investigator Responsibility | 79 |
| 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB) | 79 |
| 18.4. Informed Consent | 80 |
| 18.5. Privacy of Personal Data | 80 |
| 19. STUDY RECORD RETENTION | 82 |
| 20. FINANCIAL CONSIDERATIONS | 82 |
| 21. PUBLICATION | 83 |
| 22. REFERENCES | 83 |
| APPENDIX A : PATIENT REPORTED OUTCOMES (STUDY | |
| QUESTIONNAIRES) AND QUEST/QUANT QUESTIONNAIRES : | |
| APPENDIX B: PATIENT INSTRUCTION GUIDE | |
| APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT) | 127 |

| APPENDIX D: PRESBYOPIC SYMPTOMS QUESTIONNAIRE | 156 |
|---|---|
| APPENDIX E: OCULAR DOMINANCE | 157 |
| APPENDIX F: TEST LENS FITTING GUIDE | 158 |
| APPENDIX G: NON-INVASIVE TEAR BREAK-UP TIME (NITBUT) | 160 |
| APPENDIX H: LOGMAR VISUAL ACUITY | 161 |
| APPENDIX I: RANDOT STEREOPSIS | 162 |
| APPENDIX J: UNILATERAL COVER TEST | 163 |
| APPENDIX K: FIXATION DISPARITY | 164 |
| APPENDIX L: DISTANCE CONTRAST THRESHOLD | 165 |
| APPENDIX M: BLUR TOLERANCE TESTING | 166 |
| APPENDIX N: PERSONALITY TEST (BIG 5) | 168 |
| APPENDIX O: PRE-FIT INTERVIEW | |
| APPENDIX P: POST-FIT INTERVIEW | 170 |
| APPENDIX Q: MEASUREMENT OF LENS CENTRATION WITH MEDMONT TOPOGRAPHER | 171 |
| APPENDIX R: | 173 |
| DETERMINATION OF NEAR ADD | 174 |
| LENS FITTING CHARACTERISTICS | 182 |
| SUBJECT REPORTED OCULAR SYMPTOMS | 189 |
| DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS | 191 |
| BIOMICROSCOPY SCALE | 198 |
| KERATOMETRY PROCEDURE | 204 |
| MEASUREMENT OF COAS WAVEFRONT ABBERATIONS | 206 |
| LENS INSERTION AND REMOVAL | 214 |
| WAM-5500 ON-AXIS AUTO REFRACTION MEASUREMENT | 217 |
| Work-aid: Measuring Pupil Diameter with NeurOptics VIP-300 Variable Pupillometer | 221 |
| PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE | 225 |
| TABLE OF CONTENTS Figure 1: Study Flowchart | 23 |
| 1.5 % 1. Stady 1.10 (1.0 house) | 23 |
| TABLE OF CONTENTS | |
| Table 1: Test Article | |
| Table 2: Ancillary Supplies | |

| Table 4: Study procedures by visit | 3 | 5 |
|------------------------------------|---|---|
|------------------------------------|---|---|

#### PROTOCOL TITLE, NUMBER, VERSION

Title: Characterizing Successful Multifocal Contact Lens Wearers

Protocol Number: CR-5945 Version: 9.0 Amendment 8 Date: 20December 2019

#### SPONSOR NAME AND ADDRESS

Johnson & Johnson Vision Care (JJVC) 7500 Centurion Parkway Jacksonville, FL 32256

#### MEDICAL MONITOR



The Medical Monitor must be notified by the clinical institution/site by e-mail, fax, or telephone within 24 hours of learning of a Serious Adverse Event. The Medical Monitor may be contacted during business hours for adverse event questions. General study related questions should be directed towards your assigned clinical research associate.

The Medical Monitoring Plan is maintained as a separate document and included in the Trial Master File.

#### **AUTHORIZED SIGNATURES**

The signature below constitutes the approval of this protocol and the attachments, and provides the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable U.S. federal regulations, ICH guidelines, ISO 14155, and the Declaration of Helsinki.

| Author | | 24 Jan 2020<br>DATE |
|---|---|---|
| Reviewer | | 24 jan 2020<br>DATE |
| Study Responsible<br>Clinician | See Electronic Signature Report | DATE |
| Clinical Operations<br>Manager | See Electronic Signature Report | DATE |
| Biostatistician | See Electronic Signature Report | DATE |
| Data Management | See Electronic Signature Report | DATE |

| Reviewer | No Fellow Review Required | |
|----------|---------------------------------|------|
| | | DATE |
| Approver | See Electronic Signature Report | |
| | | DATE |

#### **CHANGE HISTORY**

| Version | Originator | Description of Change(s) and Section<br>Number(s) Affected | Date |
|---|---|---|---|
| 1.0 | | Original Protocol | 18 October 2018 |
| 2.0<br>Amendment<br>1 | | <ul> <li>PRO Spec revised in Appendix A and also combined Appendices A and B.</li> <li>Alphabetizing of Appendices updated due to Appendices A and B being combined into one document in Appendix A.</li> <li>Added the labels for primary and secondary packaging to Section 6.4 Packaging and Labeling.</li> <li>Removed the Compass lens over labelling # in Section 6.1 Identity of Test Articles.</li> <li>Table of Contents updated.</li> <li>Version and Date updated throughout the protocol.</li> </ul> | 14 November<br>2018 |
| 3.0<br>Amendment<br>2 | | <ul> <li>Appendix A-corrected spelling errors in PRO spec.</li> <li>Synopsis and section 3.3 exclusion criteria 10 added previous cataract surgery.</li> <li>Synopsis, section1 and section 4.1-replaced observational with Single-Arm. Also in 4.1 removed observational from one of the sentences.</li> <li>Section 4.2 replaced observational with exploratory.</li> <li>Version and Date updated throughout the protocol.</li> </ul> | 21 December<br>2018 |
| 4.0<br>Amendment<br>3 | | <ul> <li>Section 7.2-removed step 1.3; step 2.6 corrected appendix from L to M; section 3.5 removed the note instruction</li> <li>Section 7.3-removed steps U7-U9.</li> <li>Appendix M-updated blur tolerance procedure.</li> <li>Appendix A-updated PRO spec.</li> <li>Version and Date updated throughout the protocol.</li> </ul> | 08 February<br>2019 |

| 5.0 | | Appendix A-updated PRO spec. | 11 February |
|---|---|---|---|
| Amendment | | Version and Date updated throughout | 2019 |
| 4 | | the protocol. | 2017 |
| 6.0 | _ | Section 1.5. Removed statement | 22 February |
| Amendment | | regarding studies | 2019 |
| 5 | | not having completed CSR's as | 2019 |
| 3 | | they are now complete. | |
| | | • | |
| | - | Version and Date updated throughout | |
| 7.0 | | the protocol. | 00 M 2010 |
| 7.0 | - | Section 6.4. Removed secondary label | 09 May 2019 |
| Amendment | | and clarified how lenses will be placed | |
| 6 | | in separate clear plastic bags. | |
| | | Appendix M. Updated blur tolerance | |
| | | procedure. | |
| | 12 | Version and Date updated throughout | |
| 22,100 | 8/ 1 | the protocol. | |
| 8.0 | | Version and Date updated throughout | 21 June 2019 |
| Amendment | | the protocol. | |
| 7 | 1121 | Revised Inclusion # 8 in the Synopsis | |
| | | and section 3.2 | |
| | 19 <del>4</del> | Updated sections 1.3, 1.4 and 1.5. | |
| | 2.5 | Section 6.1- removed estimated | |
| | | number of study lenses and updated | |
| | | lens information | |
| | 100 | Added Daily Disposable as key words | |
| | | Updated Investigational product to | |
| | | etafilcon A daily disposable multifocal | |
| | | lens | |
| | - | Updated lens modality to daily | |
| | | disposable throughout protocol | |
| | 8. <del>5</del> | Changed Pupillometer model from | |
| | | VIP-200 to VIP-300 throughout | |
| | | protocol | |
| | 0- | Removed all references to Alcon Clear | |
| | | Care Solution throughout protocol | |

| | | 9 | ** | |
|---|---|---|---|---|
| 9.0 | | Ti. | Version and Date updated throughout the | 20 December |
| Amendment | | | protocol. | 2019 |
| 8 | - | - | Signature page-added degree to | |
| | | | approver | |
| | | 1-0 | Section 7.2-lenses and patient | |
| | | | instruction steps change language to | |
| | | | allow for dispensing of additional | |
| | | | lenses at the discretion of the | |
| | | | Investigator. | |
| | | | Section 14.5-removed section titled | |
| | | | Likelihood to be a successful lens wearer | |
| | | | vs. CLUE Vision Score | |
| | | | Clarified "1-meter" distance for blur test | |
| | | | throughout the protocol (as per test | |
| | | | distance in appendix M). Also in visit 2, | |
| | | | step 2.6 clarified that this test is done with | |
| | | | "intermediate (1m) refraction" | |
| | | 100 | Section 7.2-Objective accommodation: | |
| | | | added "distance" before "Sph-cyl | |
| | | | Refraction" for clarification in step 1.25. | |
| | | - | Section 7.2-Over-refraction: replaced | |
| | | | "outside of the phoropter" with "over the study CLs" in visit 2 step 2.15, and in visit | |
| | | | 3, step 3.7 | |
| | | | Section 7.2-Stereo-Acuity: clarified that | |
| | | 15.50 | Stereo-Acuity is measured with "CLs" in | |
| | | | steps 3.15, 4.8, and 6.9 in visits 3, 4 and 6, | |
| | | | respectively. | |
| | | - | Section 7.2-Contrast threshold: clarified | |
| | | | that Contrast threshold is measured with | |
| | | | "CLs" in steps 3.16, 4.9, and 6.10 in visits | |
| | | | 3, 4 and 6, respectively. | |

#### **SYNOPSIS**

| Protocol Title | Characterizing Successful Myopic Multifocal Contact Lens<br>Wearers |
|---|---|
| Sponsor | JJVC, 7500 Centurion Parkway, Jacksonville, FL 32256 |
| Clinical Phase | Development phase, Phase 0 |
| Trial Registration | This study will be registered on ClinicalTrials.gov by the |
| That Registration | sponsor. |
| Ethics approvals | Ethics approval will be sought by CORE through a |
| Etines approvais | University of Waterloo ethics committee. |
| Regulatory approval | The contact lens is approved for sale in Canada. |
| Test Article(s) | Investigational Products: Etafilcon A Multifocal Contact |
| Test TittleTe(s) | Lens |
| | Control Products: None |
| Wear and Replacement | Wear Schedule: Daily wear |
| Schedules | Replacement Schedule: Daily Disposable |
| Objectives | <b>Primary Objectives</b> : To determine if the QUEST questionnaire, collected at baseline, are significantly correlated with subject groups that are classified as being 'likely to be successful' and/or 'likely to be unsuccessful' after wearing an investigational multifocal (ML) contact lens (CL). |
| | Secondary Objectives: To determine if certain physical ocular related data is significantly correlated with subject groups that are classified as being 'likely to be successful', 'likely to be unsuccessful' after wearing an investigational multifocal contact lens. |
| | Likely to be Successful Group definition: |
| | • Completed study, AND |
| | • Investigator would recommend the study CLs, AND |
| | • The subject's response on the MRD "overall quality of |
| | vision" and "overall comfort" questions as good, very |
| | good, or excellent. |
| | Likely to be Unsuccessful Group definition: |
| | • Not meeting the definition of successful. |
| Study Endpoints | Primary endpoint(s): |
| | • Quest questionnaire classification |
| | • Likelihood to be a successful lens wearer |
| | Secondary endpoint(s): |
| | Auto-refraction & keratometry (Autorefractor) |
| | Refraction including reading addition (Phoropter) |
| | • LogMAR acuity (using VA charts): monocular & binocular; distance, near (0.4 m), intermediate (1 m) |

- Fixation Disparity (with refraction): distance, & near (40 cm)
- Blur tolerance (with refraction): binocular, 1-meter distance only
- Stereo-acuity: near (40 cm)
- Contrast threshold: OD, OS, and OU distance only
- Pupil size: Photopic; OD & OS, distance, intermediate (1 m) & near (40 cm)
- Pupil size: Scotopic; OD & OS, distance, intermediate (1 m) & near (40 cm)
- Non-invasive tear break-up time: OD & OS (Placido disc)
- Objective accommodation with distance refraction (WAM 5500: 4 m, 1 m, and 40 cm target) OD & OS
- Spherical aberration: COAS, over 2 seconds after blink, OD & OS @ distance target
- Coma
- Other higher order aberrations
- Medmont Lens centration OD and OS

#### Study Design

This is a prospective, single-arm, and bilateral dispensing study.

There will a total of 6 visits:

Visit 1 (Screening and Baseline-day 0): consent, eligibility confirmation, pre-fit interview, and evaluation assessments

Visit 2 (Baseline & dispensing-Day 0): personality test, evaluation assessments, study lens fitting, CL insertion and removal training (non-CL wearers, up to 1 additional training appointments are permitted), subjective responses to CL performance, dispensing of CL

Visit 3 (1-week follow-up, lens power optimization-Day 7±3 from Visit 2): CL power optimization, lens fit assessment, evaluation assessments

Visit 4 (2-week follow-up- Day 7±3 from Visit 3): lens fit assessment, evaluation assessments, subjective responses to CL performance

Visit 5 (6-week follow-up Day 28±6 from Visit 2-): lens fit assessment, evaluation assessments, subjective responses to CL performance

Visit 6 (12-week follow-up Day 42±6 from Visit 2-): Post-fit interview, lens fit assessment, evaluation assessments, subjective responses to CL performance

| Samula Sina | Study exit: Investigator recommendation, if applicable (study CLs suitable/not suitable to prescribe, plus investigator reasons where not suitable is indicated), exit procedures. See the flow chart at the end of the synopsis table for the schematic of the study visits and procedures of main observations (Figure 1). |
|---|---|
| Sample Size | The target is to dispense lenses to 50 presbyopic Subjects who had no experience with soft multifocal contact lens wear for >2 years; total sample size 50. Enrollment is potentially likely to be up to approximately 75 to account for screen failures. |
| Study Duration | The study is anticipated to have a duration of approximately 9 months in total, with enrollment lasting approximately 6 months. |
| Anticipated Study<br>Population | All eligible Subjects will have no experience with soft multifocal contact lenses (MF CLs) for >2 years. The study population includes previous MF CL wearers, single vision CL wearers and subjects who are neophyte to CL wear; The target is to include myopes only, with a maximum reading addition of +1.75 DS. There are no sex or race requirements. All subjects need to be in the presbyopic age group ie, ≥40 years old and with a minimum add of +0.75 D. Current MF CL wearers and current monovision wearers are not eligible. |
| Eligibility Criteria | <ol> <li>Potential Subjects must satisfy all of the following criteria to participate in the study: <ol> <li>The participant must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.</li> <li>Appear able and willing to adhere to the instructions set forth in this clinical protocol.</li> <li>Is at least 40 years of age (inclusive) at the time of screening and has full legal capacity to volunteer.</li> <li>Had a self-reported eye examination in the last two years.</li> <li>The subject must either already be wearing a presbyopic correction (e.g., reading spectacles over contact lenses, or multifocal spectacles, etc.) or respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire".</li> </ol> </li> <li>Can achieve best corrected distance monocular visual acuity of at least +0.20 logMAR and binocular visual acuity of at least +0.10 logMAR with refraction.</li> </ol> |

- 7. Have a refractive cylinder of  $\leq 1.00$  D in each eye.
- 8. Has corrected best sphere equivalent distance refraction in the range of -0.50 to -6.00 DS in each eye (vertex corrected if greater than -4.00 D).
- 9. Have a reading ADD power in the range of +0.75 D to +1.75 D (inclusive) in each eye.
- 10. Have a wearable pair of spectacles if applicable (at the discretion of the investigator) to wear when they cannot wear the study lenses

Potential Subjects who meet any of the following criteria will be excluded from participating in the study:

- 1. Participation in any contact lens or lens care clinical trial within 1 week prior to study enrollment.
- 2. Employee or immediate family member of an employee of the Centre for Ocular Research & Education listed on the study Delegation Log (e.g., Investigator, Coordinator, Technician).
- 3. Is currently pregnant or lactating, by self-report, or planning a pregnancy at the time of enrollment.
- 4. Has any known active ocular disease and/or allergies, ocular infections or other abnormalities that are known to interfere with contact lens wear (at the discretion of the investigator). This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, or corneal distortion.
- 5. Is using any topical ocular medications other than lubricating eye drops.
- 6. Known to have any infectious disease (e.g., hepatitis, tuberculosis) or a contagious immunosuppressive disease.
- 7. Have any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear (at the discretion of the investigator). This may include, but not be limited to, hyperthyroidism, recurrent herpes simplex/zoster, Sjogren's syndromes, xerophthalmia, acne rosacea, Stevens-Johnson syndromes.
- 8. Had a diagnosis of a condition known to affect ocular prescription or ocular surface or tear film e.g., rheumatoid arthritis, diabetes.
- 9. Had a change within the previous 3 months to the dosage of a systemic medication known to affect ocular prescription or ocular surface or tear film (e.g., steroids) that in the opinion of the investigator may affect a study outcome variable.

| | <ol> <li>Has undergone cataract or refractive error surgery (e.g., radial keratotomy, PRK, LASIK, etc.), or has any planned (during the study) major surgery (e.g. hip replacement), or any planned ocular surgery (e.g. cataract or refractive error surgery).</li> <li>Is a current rigid contact lens wearer, or is wearing contact lenses on extended wear basis, or has a history of extended wear in the past 6 months.</li> <li>Has worn soft MF CLs in the past 2 years or is a habitual wearer of monovision CLs.</li> <li>Has a constant unilateral strabismus at both far and near distances, or Has anisometropia &gt;2 D between both eyes, or has amblyopia.</li> <li>Has a known sensitivity to the diagnostic pharmaceuticals to be used in the study (Refresh Plus® rewetting drop solution, or Sodium Fluorescein.</li> <li>Has any Grade 3.0 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the Biomicroscopy classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate</li> </ol> |
|---|---|
| | contact lens wear (at the discretion of the investigator). |
| Disallowed Medications/Interventions | Any medications (Rx or OTC, systemic or topical) that may interfere with contact lens wear (at the discretion of the investigator). No ocular topical medications (e.g. Restasis, Xiidra, ocular steroids) except lubricating eye drops. |
| Measurements and | Visit 1 (Screening, Baseline): |
| Procedures | Subjects will attend wearing their habitual contact lenses or if not a contact lens wearer then spectacles (if applicable), they also need to bring any distance / reading spectacles, package of their CLs, lens care solution, and rewetting/lubrication eye drops to the appointment. |
| | Consent procedures |
| | Demographics, health and medication, habitual correction type, CL wearing history. |
| | Subjective responses to CL performance (CLUE questionnaire). If habitual contact lens wearers. |
| | CL experience and expectations (Quest-Quant questionnaire) |

Interview (pre-fit) to identify: Subjects' success criteria; reasons for success/failure; visual demands eg. laptop, shift work, night driving etc.

logMAR acuity with habitual contact lenses/spectacles (if applicable): monocular & binocular; distance Auto-refraction & keratometry Refraction including reading addition logMAR acuity (with refraction): monocular & binocular; distance, near (0.4 m), intermediate (1 m) Ocular dominance

Unilateral cover test: distance & near (40 cm) Stereo-acuity with refraction: near (40 cm)

Fixation Disparity: distance& near (40 cm) Contrast threshold: OD, OS, and OU distance only

Non-invasive tear break-up time: OD & OS Objective accommodation with distance refraction (WAM 5500: 4 m, 1 m, and 40 cm target) OD & OS

Spherical aberration over bare eye: COAS, 2 secs after blink, OD & OS @ distance target Coma over bare eye
Other higher order aberrations over bare eye

logMAR acuity with habitual spectacles (if applicable): monocular & binocular; distance

#### Visit 2 (Baseline, Treatment 1):

Subjects will attend wearing their habitual spectacles (if applicable)

Personality test: BIG5

logMAR acuity with refraction: monocular & binocular; distance

Blur tolerance with refraction: binocular, 1 m distance only

Pupil size: Photopic; OD & OS, distance, intermediate (1 m)

& near (40 cm)

Pupil size: Scotopic; OD & OS, distance, intermediate (1 m) & near (40 cm)

Slit Lamp Biomicroscopy

Study CL fitting

Training for CL insertion & removal and lens care (non-CL wearers, up to 1 additional separate training visit within a maximum of 2 weeks from Visit 2 is permitted)

Post-fit Market Research (MRD) questionnaire

Study CL dispense Lens fit assessment

logMAR acuity: monocular & binocular; distance, near (0.4 m), intermediate (1 m)

#### Visit 3 Follow-up 1(1-week), lens optimization:

Subjects will attend wearing study CLs

logMAR acuity with CLs: monocular & binocular; distance & near (40 cm) only

Pupil size: Photopic with CLs; OD & OS, distance, intermediate (1 m) & near (40 cm)

Pupil size: Scotopic with CLs; OD & OS, distance, intermediate (1 m) & near (40 cm)

Slit Lamp Biomicroscopy

Study CL fitting (CL power optimization) logMAR acuity with CLs: monocular & binocular; distance & near (40 cm) only

Post-fit questionnaire (MRD)

Contrast threshold: OD, OS, and OU distance only Stereo-acuity with study CLs: near (0.4 m)

Pre-lens non-invasive tear break-up time: OD & OS Objective accommodation with CLs (WAM 5500: 4 m, 1 m, and 40 cm target) OD & OS

Spherical aberration over CLs: COAS, 2 secs after blink, OD & OS @ distance target Coma over CLs Other higher order aberrations over CLs

Imaging for lens centration using Medmont Topographer, over CLs: OD, OS

Exit logMAR acuity with CLs: monocular & binocular; distance

#### Visit 4 Follow-up 2 (2-week)

Subjects will attend wearing study CLs

Subjective responses to CL performance (CLUE questionnaire).

logMAR acuity with CLs: monocular & binocular; distance, intermediate (1 m) & near (40 cm)

Contrast threshold: OD, OS, and OU distance only Stereo-acuity with study CLs: near (0.4 m)

Lens fit assessment

Pre-lens non-invasive tear break-up time: OD & OS Objective accommodation with CLs (WAM 5500: 4 m, 1 m, and 40 cm target) OD & OS

Spherical aberration over CLS: COAS, 2 secs after blink, OD & OS @ distance target Coma over CLs
Other higher order aberrations over CLs

Slit Lamp Biomicroscopy

Exit logMAR acuity with CLs: monocular & binocular; distance

#### Visit 5 Follow-up 3 (6-week):

Subjects will attend wearing study CLs

Subjective responses to CL performance (CLUE questionnaire)

logMAR acuity with CLs: monocular & binocular; distance, intermediate (1 m) & near (40 cm)

| | <del>,</del> |
|---|---|
| | Lens fit assessment |
| | Slit Lamp Biomicroscopy |
| | Exit logMAR acuity with CLs: monocular & binocular; distance |
| | Visit 6 Follow-up 4 (12-week): |
| | Interview (post-fit) Subjective responses to CL performance (CLUE questionnaire, market research questionnaire) |
| | logMAR acuity with CLs: monocular & binocular; distance, intermediate (1 m) & near (40 cm) Contrast threshold: OD, OS, and OU distance only Stereo-acuity with study CLs: near (0.4 cm) |
| | Lens fit assessment Objective accommodation with CLs (WAM 5500: 4 m, 1 m, and 40 cm target) OD & OS |
| | Spherical aberration over CLs: COAS, 2 secs after blink, OD & OS @ distance target Coma over CLs |
| | Other higher order aberrations over CLs |
| | Slit Lamp Biomicroscopy |
| | Investigator RecommendationInvestigator recommendation, if applicable (study CLs suitable/not suitable to prescribe, plus investigator reasons where not suitable is indicated) Exit Slit Lamp Biomicroscopy Exit logMAR acuity with refraction: monocular & binocular; distance. |
| | Final Evaluation |
| | Biomicroscopy (if subject is discontinued and Biomicroscopy was not completed in the Visit) |
| | PRO (CLUE and MRD) contact lens questionnaires (if subject discontinued). |
| Microbiology or Other | None |
| Laboratory Testing Study Termination | The occurrence of one or more Unanticipated Adverse<br>Device Effect (UADE), or any SAE where relationship to |
| | study agent cannot be ruled out, will result in stopping further dispensing investigational product. In the event of a |

| | UADE or SAE, the Sponsor Medical Monitor may unmask |
|---|---|
| | (if applicable) the treatment regimen of participant(s) and |
| | may discuss this with the Principal Investigator before any |
| | further Subjects are enrolled. |
| Ancillary Supplies/ Study- | No lens care solution will be used in this study. The lenses |
| Specific Materials | will be worn on a daily disposable modality. |
| Principal Investigator(s) | Prof. Lyndon Jones |
| and Study | Centre for Ocular Research and Education, University of |
| Institution(s)/Site(s) | Waterloo, CANADA |

Figure 1: Study Flowchart

## Visit 1 (Screening): Consent, eligibility confirmation, Quest questionnaire, PRO (CLUE) questionnaire for habitual CL wearers, pre-fit interview, and evaluation assessments Visit 2 (Baseline & Treatment 1): Personality test, evaluation assessments, CL fitting, CL insertion and removal training (non-CL wearers), Subjective responses to CL performance PRO (MRD) Visit 3 (Follow-up 1(1-week), lens power optimization): CL power optimization, CL fit assessment, evaluation assessments, Subjective responses to CL performance PRO (MRD) Visit 4 Follow-up 2 (2-week): Subjective responses to CL performance PRO (CLUE) CL fit assessment, evaluation assessments Visit 5 Follow-up 3 (6-week): Subjective responses to CL performance PRO (CLUE) CL fit assessment, evaluation assessments Visit 6 Follow-up 4 (12-week): Post-fit interview, lens fit assessment, evaluation assessments, Subjective responses to CL performance PRO (CLUE + MRD), study exit including Investigator's recommendation (study CLs suitable/not suitable)

#### COMMONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS

ADD Plus Power Required For Near Use

ADE Adverse Device Effect

AE Adverse Event/Adverse Experience

BCVA Best Corrected Visual Acuity

BSCVA Best Spectacle Corrected Visual Acuity

CFR Code of Federal Regulations

CI Confidence Interval

CL Contact lens

CLUE Contact Lens User Experience

COAS Complete Ophthalmic Analysis System

COM Clinical Operations Manager

CORE Centre for Ocular Research and Education

CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organization

CT Center Thickness

D Diopter

DMC Data Monitoring Committee eCRF Electronic Case Report Form EDC Electronic Data Capture

ETDRS Early Treatment Diabetic Retinopathy Study

FDA Food and Drug Administration

GCP Good Clinical Practice
HCVA High Contrast Visual Acuity

HIPAA Health Insurance Portability and Accountability Act

HIV Human Immunodeficiency Virus

IB Investigator's Brochure
ICF Informed Consent Form
ICL Informed Consent letter

ICHInternational Council on HarmonizationIDEInvestigational Device ExemptionIECIndependent Ethics CommitteeIRBInstitutional Review Board

ISO International Organization for Standardization

ITT Intent-to-Treat

JJVC Johnson & Johnson Vision Care, Inc.

LC Limbus Center

LogMAR Logarithm of Minimal Angle of Resolution MedDRA<sup>©</sup> Medical Dictionary for Regulatory Activities

MF Multifocal

MF CLs Multifocal Contact Lenses MOP Manual of Procedures NIH National Institutes of Health

NITBUT Non Invasive Tear Break Up Time

OD Right Eye

OHRP Office for Human Research Protections
OHSR Office for Human Subjects Research

OS Left Eye
OU Both Eyes

PD Protocol Deviation

PHI Protected Health Information

PI Principal Investigator
PIG Patient Instruction Guide
PQC Product Quality Complaint
PRO Patient Reported Outcome

QA Quality Assurance QC Quality Control

SAE Serious Adverse Event/Serious Adverse Experience

SAP Statistical Analysis Plan SAS Statistical Analysis System

SD Standard Deviation

SOP Standard Operating Procedure

UADE Unanticipated Adverse Device Effect

USADE Unanticipated Serious Adverse Device Effect

UW University of Waterloo

VA Visual Acuity

#### 1. INTRODUCTION AND BACKGROUND

Despite the growing number of presbyopes by aging, only a small fraction of presbyopic patients can be categorized as successful habitual soft multifocal (MF) contact lens (CL) wearers. Some habitual spectacle/single vision contact lens wearers in the presbyopic age group may have tried soft MF CLs in the past and dropped out from MF CL wear for various reasons. This single-arm study was designed to investigate the possible underlying reasons for achieving success or dropping out from soft MF CL wear.

#### 1.1. Name and Descriptions of Investigational Products

This study will test a etafilcon Multifocal CL. Further details about the test article is found in Section 6 of this protocol. No control products will be used in this study.

#### 1.2. Intended Use of Investigational Products

The intended use of the investigative product is for correcting presbyopia. During the study, the test article will be worn bilaterally in daily wear, daily disposable modality for at least 6 hours per day every day for approximately 12 weeks.

#### 1.3. Summary of Findings from Nonclinical Studies

N/A

#### 1.4. Summary of Known Risks and Benefits to Human Subjects

- This is a minimal risk study because of the use of an approved and previously marketed contact lens (1-Day Acuvue Moist brand Multifocal) and standard optometric assessments.
- Participants may not benefit directly in this study, other than having an opportunity to wear a marketed multifocal contact lens, at no cost to them. Information from this study may help the study sponsor to come up with new soft multifocal contact lens designs to help others in the future.

See package insert for additional information.

# 1.5. Relevant Literature References and Prior Clinical Data Relevant to Proposed Clinical Study

N/A.

#### 2. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES

#### 2.1. Objectives

Primary Objective(s):

To determine if the QUEST questionnaire, collected at baseline, are significantly correlated with subject groups that are classified as being 'likely to be successful' and/or 'likely to be unsuccessful' after wearing an investigational multifocal contact lens.

#### Secondary Objective(s):

To determine if certain physical ocular related data is significantly correlated with subject groups that are classified as being 'likely to be successful', 'likely to be unsuccessful' after wearing an investigational multifocal contact lens.

#### Likely to be Successful Group definition:

- Completed study, AND ...
- Investigator would recommend the study CLs, AND ...
- The subjects' response on the MRD "overall quality of vision" and "overall comfort" questions as good, very good, or excellent.

#### Likely to be Unsuccessful Group definition:

• Not meeting the definition of successful.

Exploratory Objective(s): BIG 5 Personality Assessment

#### 2.2. Endpoints

#### Primary Endpoints

- Likelihood to be a successful lens wearer \*
- Quest questionnaire classification

#### Secondary Endpoints

- Auto-refraction & keratometry (Autorefractor)
- Refraction including reading addition (Phoropter)
- LogMAR acuity (using VA charts): monocular & binocular; distance, near (0.4 m), intermediate (1 m)
- Fixation Disparity (with refraction): distance, & near (40 cm)
- Blur tolerance (with refraction): binocular, 1-meter distance only
- Stereo-acuity: near (40 cm)
- Contrast threshold: OD. OS, and OU distance only
- Pupil size: Photopic; OD & OS, distance, intermediate (1 m) & near (40 cm)
- Pupil size: Scotopic; OD & OS, distance, intermediate (1 m) & near (40 cm)
- Non-invasive tear break-up time: OD & OS (Placido disc)
- Objective accommodation with distance refraction (WAM 5500: 4 m, 1 m, and 40 cm target) OD & OS
- Spherical aberration: COAS, 2 secs after blink, OD & OS @ distance target
- Coma
- Other higher order aberrations
- Lens centration OD & OS: Medmont

#### Exploratory Endpoint(s):

- BIG 5 Personality Assessment
- CLUE and Market Research Questionnaires

#### \*Likely to be Successful Group definition:

- Completed all required study visits, AND ...
- Investigator would recommend the study CLs, AND ...
- The subjects' response on the MRD "overall quality of vision" and "overall comfort" questions as good, very good or excellent.

#### Likely to be Unsuccessful Group definition:

• Not meeting the definition of successful.

#### 2.3. Hypotheses

#### Primary Hypothesis

• At least 75% of the subjects who are classified by Quest questionnaire as being "discontented and driven" will be in the "likely to be successful" group. The Quest questionnaire will be collected at baseline.

#### Secondary Hypothesis

• At least one of the secondary endpoints will be significantly correlated with the success classification of the subjects after adjusting for age, sex and ADD power.

#### 3. TARGETED STUDY POPULATION

#### 3.1. General Characteristics

There are no sex or race requirements for potential study Subjects.

All Subjects need to be in the presbyopic age group i.e. 40 years or older and with a minimum add of +0.75 D. All eligible Subjects will have no experience with soft multifocal lenses (MF CLs) for >2 years. The study population includes previous MF CL wearers, Single vision CL wearers and Subjects who are neophyte to CL wear. Current MF CL wearers and current monovision wearers are not eligible.

The study will include myopes only, with reading ADDs from +0.75 up to and including +1.75 DS.

#### 3.2. Inclusion Criteria

Potential Subjects must satisfy all of the following criteria to be enrolled in the study:

- 1. The participant must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
- 2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
- 3. Is at least 40 years of age (inclusive) at the time of screening and has full legal capacity to volunteer.
- 4. Had a self-reported eye examination in the last two years.
- 5. The subject must either already be wearing a presbyopic correction (e.g., reading spectacles over contact lenses, or multifocal spectacles, etc.) or respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire".

- 6. Can achieve best corrected distance monocular visual acuity of at least +0.20 logMAR and binocular visual acuity of at least +0.10 logMAR with refraction.
- 7. Have a refractive cylinder of  $\leq 1.00$  D in each eye.
- 8. Has corrected best sphere equivalent distance refraction in the range -0.50 D of -6.00 D in each eye (vertex corrected if greater than -4.00D).
- 9. Have a reading ADD power in the range of +0.75 D to +1.75 D (inclusive) in each eye.
- 10. Have a wearable pair of spectacles (at the discretion of the investigator) to wear when they cannot wear the study lenses.

#### 3.3. Exclusion Criteria

Potential Subjects who meet any of the following criteria will be excluded from participating in the study:

- 1. Participation in any contact lens or lens care clinical trial within 1 week prior to study enrollment.
- 2. Employee or immediate family member of an employee of the Centre for Ocular Research & Education listed on the study Delegation Log (e.g., Investigator, Coordinator, Technician).
- 3. Is currently pregnant or lactating, by self-report, or planning a pregnancy at the time of enrollment.
- 4. Has any known active ocular disease and/or allergies, ocular infections or other abnormalities that are known to interfere with contact lens wear (at the discretion of the investigator). This may include, but not be limited to entropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, or corneal distortion.
- 5. Is using any topical ocular medications other than lubricating eye drops.
- 6. Known to have any infectious disease (e.g., hepatitis, tuberculosis) or a contagious immunosuppressive disease.
- 7. Have any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear (at the discretion of the investigator). This may include, but not be limited to, hyperthyroidism, recurrent herpes simplex/zoster, Sjogren's syndromes, xerophthalmia, acne rosacea, Stevens-Johnson syndromes.
- 8. Had a diagnosis of a condition known to affect ocular prescription or ocular surface or tear film e.g., rheumatoid arthritis, diabetes.
- 9. Had a change within the previous 3 months to the dosage of a systemic medication known to affect ocular prescription or ocular surface or tear film (e.g., steroids) that in the opinion of the investigator may affect a study outcome variable.
- 10. Has undergone cataract or refractive error surgery (e.g., radial keratotomy, PRK, LASIK, etc.), or has any planned (during the study) major surgery (e.g., hip replacement), or any planned ocular surgery (e.g., cataract or refractive error surgery).
- 11. Is a current rigid contact lens wearer, or is wearing contact lenses on extended wear basis, or has a history of extended wear in the past 6 months.
- 12. Has worn soft MF CLs in the past 2 years or is a habitual wearer of monovision CLs.
- 13. Has a constant unilateral strabismus at both far and near distances, or has anisometropia >2 D between both eyes, or has amblyopia.

- 14. Has a known sensitivity to the diagnostic pharmaceuticals to be used in the study (Refresh Plus®rewetting drop solution, or Sodium Fluorescein).
- 15. Has any Grade 3.0 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the biomicroscopy classification scale, any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear (at the discretion of the investigator).

#### 3.4. Enrollment Strategy

All Subjects need to be in the presbyopic age group ie.  $\geq$ 40 years old and with a minimum add of +0.75 D. There are no sex or race requirements.

All eligible Subjects will have no experience with soft multifocal lenses (MF CLs) for >2 years. The study population includes previous MF CL wearers, Single vision CL wearers and Subjects who are neophyte to CL wear. Current MF CL wearers and current monovision wearers are not eligible.

The study will include myopes only, with reading ADDs from +0.75 up to and including +1.75 DS.

#### 4. STUDY DESIGN AND RATIONALE

#### 4.1. Description of Study Design

This will be a prospective, single group, single-arm, and bilateral dispensing study. There will be no randomization and no masking in this non-controlled single-arm study. There also will be no wash out period. Subjects will be assigned to a single study lens type to be worn bilaterally in daily wear, and daily disposable modality, for at least 6 hours per day every day for approximately 12 weeks.

There will 6 visits in this study:

Visit 1: screening and baseline; eligibility confirmation, Quest questionnaire, pre-fit interview

Visit 2: baseline; personality test, study lens fitting

Visit 3: 1-week; CL power optimization

Visit 4: 2-week assessments with study CLs

Visit 5: 6-week assessments with study CLs

Visit 6: 12-week assessments with study CLs, post-fit interview

#### 4.2. Study Design Rationale

This study was designed based on its exploratory nature. The single-arm design is used to explore differences in personality and qualitative interview variations as well as differences in refraction and anatomical measurements between successful and unsuccessful Subjects with study soft multifocal lenses.

#### 4.3. Enrollment Target and Study Duration

- Up to approximately 75 Subjects will be screened, with a target of dispensing product to up to 50 subjects who may complete the study. Subjects will be recruited using CORE records and advertising approved by the University of Waterloo (UW) Office of Research Ethics (ORE).
- Point of enrollment in this study will be execution of informed consent.
- There will be a total of 6 study visits including the study screening visit during which consent, eligibility confirmation, interview and evaluation assessments will be conducted.
- The study will last approximately 9 months and include a 6 month enrollment period.
- This will be a single site study. Study visits will be conducted at Centre for Ocular Research & Education (CORE), University of Waterloo, Ontario.

#### 5. TEST ARTICLE ALLOCATION AND MASKING

#### 5.1. Test Article Allocation

There will be no randomization in this single arm study as there will be no controls, and only one test article is used.

#### 5.2. Masking

Not applicable. There will be no masking in this study.

Subjects who are discontinued will not be replaced.

#### 5.3. Procedures for Maintaining and Breaking the Masking

Not applicable. There will be no masking in this study.

#### 6. STUDY INTERVENTION

#### 6.1. Identity of Test Articles

The following contact lens will be used in this study:

Table 1: Test Article

| | Test Article |
|--------------------------------------|----------------------------|
| Name | Acuvue® Moist Multifocal |
| | Contact Lens |
| Manufacturer | Johnson & Johnson® Vision |
| | Care, Inc. |
| Health Canada License | #2519 |
| Compass Protocol(s) and/or Lot | Secondary package will be |
| Number or Other Identifier | labeled |
| Lens Material | etafilcon A |
| Nominal Base Curve @ 22°C | 8.4 mm |
| Nominal Diameter @ 22°C | 14.3 mm |
| Nominal Distance Powers (D) | Plano to -6.00 D in 0.25 D |
| pa sour | steps |
| Nominal ADD Powers (D) | Low, Mid, High |
| Water Content (Optional) | 58% |
| Center Thickness (Optional) | 0.084 mm (-3.00 D) |
| Oxygen Permeability (Dk) | 28.0 |
| Wear Schedule in Current Study | Daily Wear |
| Replacement Frequency | Daily Disposable |
| Packaging Form (vial, blister, etc.) | Blister |

#### 6.2. Ancillary Supplies/Products

The following rewetting drop will be used in this study:

Table 2: Ancillary Supplies

| Solution | Refresh Plus® Rewetting |
|------------------|-------------------------|
| Name/Description | Drops |
| Manufacturer | Allergan |
| Preservative | Non-preserved |
| Active agent | N/A |
| DIN# | 02049260 |

#### 6.3. Administration of Test Articles

Test articles will be dispensed to participants meeting all eligibility requirements, including any dispensing requirements set forth in this clinical protocol. Subjects will be dispensed an

adequate supply of test articles to complete the study. Lost or damaged test articles may be replaced at the discretion of the Investigator and/or the Sponsor.

#### 6.4. Packaging and Labeling

The test articles will be packaged in blisters as the primary packaging.

The test articles will be in labeled cartons based upon their lens power. The sample label is shown below:

# Sponsored By/Parrainé par: Johnson & Johnson Vision Care, Inc. 7500 Centurion Parkway Jacksonville, FL 32256, USA For Use in Clinical Study Destinée à l'étude clinique Not for Sale Ne peut être vendu

#### 6.5. Storage Conditions

Test articles will be maintained at ambient temperatures at the clinical site. Test articles must be kept under secure conditions.

#### **6.6.** Collection and Storage of Samples

When possible, any lens or test article associated with an Adverse Events and/or a Product Quality Complaint must be retained and stored in a glass vial with moderate solution pending directions from the sponsor for potential return back to JJVC.

#### 6.7. Accountability of Test Articles

JJVC will provide the Investigator with sufficient quantities of study articles and supplies to complete the investigation. The Investigator is asked to retain all lens shipment documentation for the test article accountability records.

Test article must be kept in a locked storage cabinet, accessible only to those assigned by the Investigator for dispensing. The Investigator may delegate this activity to authorized study site personnel listed on the Site Delegation Log. All test articles must be accounted. This includes:

- 1. What was dispensed for the participant for trial fitting, to wear out of the office, or issued for the participant to replace appropriately between visits
- 2. What was returned to the Investigator unused
- 3. The number and reason for unplanned replacements.

The Investigator will collect all unused test articles from the Subjects at the end of the participant's participation, when possible. Subject returned unused test articles must be separated from the clinical study inventory of un-dispensed test articles and must be labeled

with the participant number and date of return. Following final reconciliation of test articles by the monitor, the Investigator or monitor will return/destroy all unused test articles to JJVC.

If there is a discrepancy between the shipment documents and the contents, contact the study monitor <u>immediately.</u>

#### 7. STUDY EVALUATIONS

#### 7.1. Time and Event Schedule

There will be 6 study visits including the screening, interview and study assessments.

Table 3: Time and Events

| Visit 1: Screening and Baseline 1 | Day 0 |
|------------------------------------------|------------------------|
| Visit 2: Baseline 2 & Dispense | Day 0 |
| Visit 3: 1-week follow-up & optimization | Day 7± 3 days from V2 |
| Visit 4: 2-week follow-up | Day 7± 3 days from V3 |
| Visit 5: 6-week follow-up | Day 28± 6 days from V4 |
| Visit 6: 12-week follow-up | Day 42± 6 days from V5 |

<sup>\*</sup>Note: An additional insertion and removal visit may occur after Visit 2 if required for additional training.

#### 7.1.1. Additional screening visits

No additional screening visits will be allowed.

#### 7.2. Detailed Study Procedures

There will be a total of 6 study visits including a screening and baseline visit in this study. The investigator will determine participant eligibility using the inclusion and exclusion criteria. Ineligible Subjects will be discontinued from the study.

All Subjects will attend the study screening visits wearing their habitual spectacles. They will attend the rest of the study visits (3-6) after at least 2 hours of study MF CL wear.

The study procedures per visit are listed in the Table 4 below, with more detailed information provided afterwards. All Subjects will undergo all procedures except for CL insertion/removal training, which is not applicable to habitual CL wearers. One additional separate training session within maximum of 2 weeks from Visit 2 is permitted in the study.

Table 4: Study procedures by visit

| Visit Information | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Final |
|---|---|---|---|---|---|---|---|
| VISIT IIIOIIIIAUOII | Screening | Baseline, | 1-week | 2-week | 6-week | 12- | Evaluation |
| | Baseline | personality | Follow-up | Follow- | Follow- | week | Evaluation |
| | Pre-fit | test, lens | 1, | up 2 | up 3 | Follow- | |
| | interview | fitting & | CL power | up 2 | up 3 | up 4 | |
| | merview | training | optimizatio | | | up 4 | |
| | | lraining | n | | | | |
| Time Point | Day 0 | Day 0 | Week 1 | Week 2 | Week 6 | Week 1 | |
| THE COLOR CONTROL CONTROL CONTROL | | (1-14 days | Day 7± 3 | Day 7± | Day 28± | 2 | |
| | | V1) | from V2 | 3 from | 6 from | Day 42 | |
| | | 10/20- | 0.04.04.04.04.04.04.04.04.04.04.04.04.04 | V3 | V4 | ±6 from | |
| | | | | 19000 | 34. 36 | V5 | |
| Estimated Visit | 3.5 hrs | 3.5 hrs | 2.5 hrs | 2.5 hrs | 1 hr | 2.5 hrs | 0.5 hr |
| Duration | 5-000 LL 180-50-781 | . 15-40-00-00-00-00-00-00-00-00-00-00-00-00- | | | | | |
| Statement of | | | | | | | |
| Informed Consent | X | | | | | | |
| Demographics | X | | | | | | |
| Medical | | | | | | | |
| History/Concomita | | | | | | | |
| nt Medications | X | | | | | | |
| Adverse Event and | | | | | | | |
| Concomitant | | | | | | | |
| Medications | | | | | | | |
| Review | X | X | X | X | X | X | |
| Habitual visual | | | | | | | |
| correction | | | | | | | |
| information | X | | | | | | |
| Contact Lens wear | | | | | | | |
| history | X | | | | | | |
| CL experience and | | | | | | | |
| expectations | | | | | | | |
| (Quest-Quant | 37 | | | | | | |
| questionnaire) | X | | | | | | |
| Interview (Pre-fit) | X | | | <u>/</u> | | | v |
| Interview (Post-fit) | | | | | | | X |
| Personality test:<br>BIG5 | | X | | | | | |
| Entrance distance | | Λ | | | | | |
| VA (spectacles) If | | | | | | | |
| applicable | X | X | | | | | |
| Entrance VA (CLs) | (2 A) | | X | X | X | X | |
| Blur tolerance with | | | | | | | |
| refraction: | | | | | | | |
| binocular, 1-meter | | | | | | | |
| distance only | | X | | | | | |
| Pupil size: | | | | | | | |
| Photopic; OD & | | | | | | | |
| OS, distance, | | | | | | | |
| intermediate (1 m) | | | | | | | |
| & near (40 cm) | | | | | | | |
| Pupil size: | | | | | | | |
| Scotopic; OD & | | X | | | | | |

| OS, distance, | | | | | | | |
|----------------------|----|---|----|----|---|-----|---|
| intermediate (1 m) | | | | | | | |
| & near (40 cm), | | | | | | | |
| with refraction | | | | | | | |
| Pupil size | | | | | | | |
| Photopic; OD & | | | | | | | |
| OS, distance, | | | | | | | |
| intermediate (1 m) | | | | | | | |
| & near (40 cm) | | | | | | | |
| Pupil size: | | | | | | | |
| Scotopic; OD & | | | | | | | |
| OS, distance, | | | | | | | |
| intermediate (1 m) | | | | | | | |
| & near (40 cm) | | | | | | | |
| with CLs | | | X | | | | |
| Auto-refraction & | | | | | | | |
| keratometry | X | | | | | | |
| Subjective Sphero- | | | | | | | |
| Cylindrical | | | | | | | |
| Refraction | X | | | | | | X |
| Reading addition | X | | | | | | |
| logMAR acuity: | | | | | | | |
| monocular & | | | | | | | |
| binocular; distance, | | | | | | | |
| near (0.4 m), | | | | | | | |
| intermediate (1 m), | | | | | | | |
| with refraction | X | | | | | | |
| logMAR acuity: | | | | | | | |
| monocular & | | | | | | | |
| binocular; distance | | | | | | | |
| & near (0.4 m) | | | | | | | |
| only, | | | | | | | |
| with CLs | | X | X | | | | |
| logMAR acuity: | | | | | | | |
| monocular & | | | | | | | |
| binocular; distance | | | | | | | |
| & near (0.4 m) | | | | | | | |
| only, | | | | | | | |
| with over- | | | | | | | |
| refraction | | X | X | | | | |
| logMAR acuity: | | | | | | | |
| monocular & | | | | | | | |
| binocular; distance, | | | | | | | |
| near (0.4 m), | | | | | | | |
| intermediate (1 m), | | | | | | | |
| with CLs | | | | X | X | X | |
| Ocular dominance | X | | | | | | |
| Unilateral cover | | | | | | | |
| test: distance & | | | | | | | |
| near (40 cm) | X | | | | | | |
| Stereo-acuity: near | | | | | | | |
| (40 cm), with near | 37 | | | | | | |
| refraction | X | | | | | | |
| Stereo-acuity: near | | | 37 | 37 | | 3.7 | |
| (40 cm), with CLs | | | X | X | | X | |
| Fixation Disparity | | | | | | | |
|---------------------|--------------|---|---|---|---|---|-----------|
| with refraction | X | | | | | | |
| Contrast threshold: | | | | | | | |
| OD, OS and OU | | | | | | | |
| distance only, | | | | | | | |
| with refraction | X | | | | | | |
| Contrast threshold: | | | | | | | |
| OD, OS and OU | | | | | | | |
| distance only, | | | | | | | |
| with CLs | | | X | X | | X | |
| Non-invasive tear | | | | | | | |
| break-up time: OD | | | | | | | |
| & OS, | | | | | | | |
| over bare eye | X | | | | | | |
| Pre-lens Non- | 71 | | | | | | |
| invasive tear | | | | | | | |
| break-up time: OD | | | | | | | |
| & OS, | | | | | | | |
| | | | v | v | | | |
| over CLs | | | X | X | | | V (:c |
| Slit Lamp | $\mathbf{v}$ | v | v | v | v | v | X (if |
| Biomicroscopy, | X | X | X | X | X | X | required) |
| Objective | | | | | | | |
| accommodation | | | | | | | |
| (WAM 5500: 4 m, | | | | | | | |
| 1 m, and 40 cm | | | | | | | |
| target) OD & OS, | | | | | | | |
| with distance | | | | | | | |
| refraction | X | | | | | | |
| Objective | | | | | | | |
| accommodation | | | | | | | |
| (WAM 5500: 4 m, | | | | | | | |
| 1 m, and 40 cm | | | | | | | |
| target) OD & OS, | | | | | | | |
| with CLs | | | X | X | | X | |
| Spherical | | | | | | | |
| aberration: COAS, | | | | | | | |
| over 2 secs after | | | | | | | |
| blink, OD & OS @ | | | | | | | |
| distance target | | | | | | | |
| Coma Other higher | | | | | | | |
| order aberrations, | | | | | | | |
| over bare eye | X | | | | | | |
| Spherical | | | | | | | |
| aberration: COAS, | | | | | | | |
| over 2 secs after | | | | | | | |
| blink, OD & OS @ | | | | | | | |
| distance target | | | | | | | |
| Coma Other higher | | | | | | | |
| order aberrations, | | | | | | | |
| over CLS | | | X | X | | X | |
| Baseline imaging | | | | | | | |
| for lens centration | | | | | | | |
| OD & OS: | | | | | | | |
| Medmont, | | | | | | | |
| over bare eye | X | | | | | | |
| | _ | | 1 | 1 | 1 | • | 1 |

| | | 1 | | | | | |
|--------------------|----------|----|-------------|-----|-----|----|---|
| Imaging for lens | | | | | | | |
| centration OD & | | | | | | | |
| OS: Medmont, | | | | | | | |
| over CLs | | | X | | | | |
| Exit distance VA | | | | | | | |
| with spectacles/ | | | | | | | |
| refraction | X | | | | | | X |
| Exit distance VA | | | | | | | |
| with CLs | | X | X | X | X | | |
| Lens Selection | | | X (if | | | | |
| Lens selection | | X | modified) | | | | |
| Lens Insertion & | | 71 | X (if | | | | |
| Settling | | X | modified) | | | | |
| Lens Power | | Λ | illoullicu) | | | | |
| Modification (if | | | | | | | |
| | | v | v | | | | |
| applicable) | | X | X | | | | |
| Subject Reported | | 37 | 37 | 3.7 | 37 | 37 | |
| Ocular Symptoms | | X | X | X | X | X | |
| Subjective | | | | | | | |
| responses to CL | | | | | | | |
| performance | | | | | | | |
| (CLUE) | X | | | X | X | X | X |
| Subjective | | | | | | | |
| responses to CL | | | | | | | |
| performance | | | | | | | |
| (market research) | | X | X | | | | |
| Lens Fit | | | | | | | |
| Assessment | | X | X | X | X | X | |
| Training for CL | | | | | | | |
| insertion & | | | | | | | |
| removal and lens | | | | | | | |
| care (non-CL | | | | | | | |
| wearers) | | X | | | | | |
| | | X | X | X | X | | |
| Study CL dispense | | Λ | Λ | Λ | Λ | | |
| Dispense Patient | | v | | | | | |
| Instruction Guide | | X | | | | | |
| Lens wear | | | 37 | 37 | 3.7 | 37 | |
| Compliance | | | X | X | X | X | |
| Study Completion | | | | | | X | |
| Investigator | | | | | | | |
| recommendation, if | | | | | | | |
| applicable (study | | | | | | | |
| CLs suitable/not | | | | | | | |
| suitable to | | | | | | | |
| prescribe, plus | | | | | | | |
| investigator | | | | | | | |
| reasons where not | | | | | | | |
| suitable is | | | | | | | |
| indicated) | | | | | | | X |
| Final Evaluation | | | | | | | X |
| | <u> </u> | 1 | | 1 | 1 | 1 | _ |

Detailed study procedures at each visit are listed below:

## VISIT 1

The Subjects must present to Visit 1 wearing habitual contact lens or if not a contact lens wearer their spectacles (if applicable). If the subject is a habitual contact lens wearer and does not have their contact lenses they must be rescheduled.

Subjects will also will be requested to bring any distance/reading spectacles, package of their CLs, lens care solution, and rewetting/lubrication eye drops to the appointment, if not they must be rescheduled.

| | | Visit 1: Screening | 4 |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.1 | Statement of<br>Informed Consent | Each participant must read, understand, and sign the Statement of Informed Consent before being enrolled into the study. The Principal Investigator or his/her designee conducting the informed consent discussion must also sign the consent form. Note: The participant must be provided a signed copy of this document. | |
| 1.2 | Demographics | Record the participant's date of birth, sex, race and ethnicity. | |
| 1.3 | Medical History<br>and Concomitant<br>Medications | Questions regarding the Subjects' medical history and concomitant medications. | |
| 1.4 | Presbyopic<br>Symptom<br>Questionnaire | Confirm the subject is either already wearing a presbyopic correction (e.g., reading spectacles over contact lenses, or multifocal spectacles, etc.) or responds positively to at least one symptom on the "Presbyopic Symptoms Questionnaire. | |
| 1.5 | Habitual Visual<br>Correction | Questions regarding the participant's habitual<br>lens/correction type and parameters. All Subjects<br>will be asked about their previous CL wear<br>including history of MF CL wear | |
| | | Interview (Pre-fit) | |
| 1.6 | CL Wear History,<br>Occupation<br>Hobbies, Visual<br>Demands, Contact<br>lens Success,<br>Reasons for<br>Success / Failure | Questions regarding the participant's: Habitual correction Occupation and hobbies Visual demands, eg laptop, shift work, night driving, etc. Success criteria with multifocal contact lenses Factors affecting success/failure with multifocal contact lenses | |

| 1.7 | Screening | All responses to Screening Inclusion Criteria | 10 |
|---|---|---|---|
| | Eligibility | questions must be answered "yes" and all | |
| | | responses to Exclusion Criteria must be answered | |
| | | "no" for the subject to be considered eligible. | |
| | | If subject is deemed to be ineligible after screening, proceed to Final Evaluation and complete Subject Disposition. Refraction and Biomicroscopy forms are not required. | |

| 6 | Visit 1: Baseline | | |
|---|---|---|---|
| Step | Procedure | Details | r 7 |
| 1.8 | Entrance Distance<br>VA (spectacles) if<br>applicable | Record distance logMAR high contrast VA with the participant's spectacles (if applicable): OD, OS, OU. Note: The acuity will be recorded to the nearest letter OD, OS, and OU. | |
| 1.9 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. | 9 |
| 1.10 | Quest-Quant<br>Questionnaire | The subject will respond to the Quest-Quant Questionnaire. | |
| 1.11 | PRO (CLUE) Questionnaire (if applicable) | If Subjects are habitual contact lens wearers they will complete the PRO (CLUE) Contact Lens performance questionnaires. | |
| 1.12 | Auto-refraction &<br>Keratometry | Record auto refraction and Keratometry results. | |
| 1.13 | Subjective Sphero-<br>Cylindrical<br>Refraction | Conduct balanced subjective Best Spherocylindrical Refraction. Record the refraction and distance logMAR visual acuity to the nearest letter. Note: Best distance monocular visual acuity with sphero-cylindrical refraction must be at least +0.20 logMAR and binocular visual acuity of at least +0.10 logMAR with refraction for the subject to enroll in the study. | |
| 1.14 | Near Add<br>Determination | The near reading addition will be determined using the binocular crossed cylinder technique at 40 cm followed by optimization in a trial frame in step 1.20 below. | |
| 1.15 | Ocular Dominance | Determine ocular dominance | |

| 1.16 | ADD Refinement | Place the BCC result in the trial frame and refine | |
|---|---|---|---|
| | | the near prescription with trial lenses (or flippers) | * |
| | | under binocular conditions. | |
| 1.17 | Near Visual | Measure Near logMAR at 40cm with near | |
| | Acuity | prescription in a trial frame. Record the near visual | |
| | | acuity OD, OS and OU. | |
| 1.18 | Unilateral Cover | Record presence/absence of strabismus in each eye | |
| | Test | (OD, OS) at distance with the Sph-cyl Refraction | |
| | | in Trial Frame. | |
| | | Then record presence/absence of strabismus in | |
| | | each eye (OD, OS) at near (40 cm) with the Sph- | |
| | | cyl Refraction and Near Add in Trial Frame. | |
| 1.19 | Biomicroscopy | Non-dilated Slit Lamp Biomicroscopy will be | |
| | 15 | performed. If the clearance of the fluorescein | · |
| | | needs to be expedited, preservative-free rewetting | |
| | | drops or saline may be instilled. | |
| | *************************************** | | |
| 1.20 | Eligibility | All responses to corresponding Screening Inclusion | |
| | | Criteria questions must be answered "yes" and all | |
| | | responses to corresponding Exclusion Criteria must | |
| | | be answered "no" for the participant to be | |
| | | considered eligible. | |
| | | If participant is deemed to be ineligible after | |
| | | baseline, proceed to Final Evaluation and | |
| | | complete Subject Disposition. Biomicroscopy and | |
| | | Sph-cyl Refraction forms are not required. | |
| 1.21 | Near Stereo-acuity | Record Stereo-acuity at 40 cm using Near Stereo- | |
| | (40 cm) | Acuity test with the Sph-cyl Refraction and Near | · · |
| | NOTES TO SEE STATE | Add in Trial Frame. | |
| 1.22 | Fixation Disparity | Record distance fixation disparity with the Sph-cyl | <u> </u> |
| | | Refraction in place. | |
| | | Then record near (40 cm) fixation disparity with | |
| | | the Sph-cyl Refraction and Near Add in Trial | |
| | | Frame. | |
| 1.23 | Contrast Threshold | Record distance contrast threshold with the Sph-cyl | |
| 1.23 | Condust Threshold | Refraction in a trial frame: OD, OS and OU. | |
| 1.24 | Tear Break-Up | Measure and record (NITBUT) OD & OS with | |
| | Time | Placido disc topographer projecting onto tear film. | |
| | (bare eye) | | 20-20 |
| 1.25 | Objective | Record objective accommodation using WAM | |
| | Accommodation | 5500 refractometer for 4m, 1m, and 40cm targets | · · |
| | | with the distance Sph-cyl Refraction OD & OS in | |

| | | Trial Frame. Record the average measurement for each distance OD, OS. |
|---|---|---|
| 1.26 | COAS<br>(bare eye) | Measure the ocular aberrations using COAS 2 secs after blink, OD & OS @ distance target Coma over bare OD, OS. |
| 1.27 | Topographer (bare eye) | Baseline imaging for lens centration using<br>Medmont Topographer, over bare eye: OD, OS |
| 1.28 | Exit distance VA | Record distance logMAR HCVA with the participant's spectacles (if applicable): OD, OS, OU. |
| 1.29 | Schedule<br>Follow-up | The subject will be scheduled to return for their next appointment in 1 to 14 days. |

The Subjects must present to Visit 2 wearing spectacles (if applicable), not having worn any contact lenses (if applicable) on the day of the visit. If the subject is wearing or has worn their lenses the day of the visit they must be rescheduled.

| | Visit 2: Baseline Treatment 1 | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 2.1. | Adverse Events<br>and Concomitant<br>Medications<br>Review | Record any changes in concomitant medications and any adverse events that may have occurred since the last scheduled study visit. | |
| 2.2. | Non-Contact Lens<br>Wear Compliance | Confirm the Subject has not worn contact lenses prior to the visit. | |
| 2.3. | Subject Reported<br>Ocular Symptoms | If the participant reports ocular symptoms with<br>their lenses, they will be recorded in the Subject<br>Reported Ocular Symptoms eCRF | |
| 2.4. | Personality test:<br>BIG5 | Have the subject conduct the personality test and record the subject's score. | |
| 2.5. | Entrance Distance<br>VA (spectacles) if<br>applicable | Record distance logMAR high contrast VA with the participant's spectacles (if applicable): OD, OS, OU. | |
| 2.6. | Blur Tolerance | Record the 1-meter distance binocular blur tolerance with intermediate (1m) refraction. | 2 |
| 2.7. | Pupil size | Measure and record pupil size in photopic & scotopic lighting using Pupilometer. Measure OD and OS at distance, intermediate(1m) and near (40cm). | |
| 2.8. | Biomicroscopy | Non-dilated Slit Lamp Biomicroscopy will be performed. | |

| | | If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. |
|---|---|---|
| 2.9. | Continuance | Confirm the participant meets the criteria to continue. |

| | Visit 2: Treatment 1 Lens Fitting | |
|---|---|---|
| Step | Procedure | Details |
| 2.10. | Lens Selection | Select the lens distance spherical equivalent power and ADD based upon the fitting guide. Record the test lens parameters (power and lot number). Place the lenses on their eyes. |
| | | Note: If a participant requires a study lens power that is not available, either as the initial selection or during a modification, they will be discontinued from the study. Complete the exit slit-lamp and VA and Final Evaluation. Sph-cyl Refraction form is not required. |
| 2.11. | Lens Insertion | Subjects or Investigator will insert the lenses. If<br>the lens is uncomfortable, inspect for damage and<br>remove, reinsert or replace as necessary. |
| | | Damaged lenses will be stored in labeled vial with<br>sterile saline, and clearly differentiated from the<br>other worn lenses that will be shipped back to the<br>Sponsor. Complete the Quality Product Complaint<br>form. |
| | Lens Settling | Allow the lenses to settle for at least 10 minutes. |
| 2.13. | Determine Visual<br>Satisfaction | Determine if the participant's vision is acceptable with the lenses. Allow the participant to look down a hallway or out of a window for distance vision assessments, and for them to read a book, magazine or similar for near vision. |
| 2.14. | logMAR HCVA<br>Acuity | Record distance and near (40cm) logMAR HCVA with study CLs: OD, OS, OU to the nearest letter |
| 2.15. | Over-refraction | Perform a distance over-refraction OD and OS using loose lenses over CLs under ambient room illumination. The distance over-refraction may also be refined under binocular conditions. Record the results. The results of the distance over-refraction may also be checked for the impact |

| | | 10-10-1 Kiel No (1879 NATE 1886 W |
|---|---|---|
| | | on near vision under monocular and/or binocular conditions. |
| 2.16. | Modifications | If the subject's vision is unacceptable for at least one distance or the Investigator determines that the visual acuity or over-refraction are not acceptable then a lens modification must be made. Up to two attempts at lens optimization are permitted if necessary, in order to achieve an acceptable distance and near binocular performance for the participant, and to enable them to wear the study lenses. Follow the fitting guide and repeat steps 2.10 to 2.15 allowing for adequate settling time between lens changes. |
| 2.17. | Lens Fit<br>Assessment | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). |
| | | <ul> <li>The subject should not proceed to wear the lenses if any of the following is observed:</li> <li>presence of limbal exposure (appearance of clear cornea) in any gaze</li> <li>presence of edge lift</li> <li>presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up).</li> </ul> |
| | | If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form. |
| 2.18. | Subject Reported<br>Ocular Symptoms | If the participant reports ocular symptoms with the lenses, they will be recorded in the Subject Reported Ocular Symptoms eCRF |
| 2.19. | Post-Fit PRO<br>(MRD)<br>Questionnaire | Subjects will complete the PRO (MRD) Contact lens performance questionnaire. |
| 2.20. | Insertion &<br>Removal Training<br>(if applicable) | Neophytes and / or lapsed wearers who the investigator determines I/R training is required will receive training on lens insertion, lens removal, lens care and general contact lens safety information. Additional lenses may be used if necessary to complete the I&R training. Record the lens information on the Lens log and in EDC. |

| | | T |
|---|---|---|
| 2.21. | Continuance<br>(Neophytes and/ or<br>lapsed wearers) | The investigator will confirm the participant is able to insert/remove study CLs independently and willing to follow lens handling and care instructions. |
| | | Note: If the subject is unable to insert and remove the contact lenses independently the subject may return for one additional visit to repeat the I/R training and be dispensed lenses if training is successful. If the subject needs additional training they will not be dispensed any lenses at this visit and will have exit visual exit visual acuity as described in step 2.22 below measured with their habitual spectacles. They will have a separate I/R training visit within two weeks and at the visit VA will be measured at distance OD, OS and OU with their habitual spectacles, biomicroscopy will be performed prior to I/R training and if the subject is successful a lens fit assessment will be performed and steps 2.22 through 2.27 below will be repeated. If unsuccessful the subject will be discontinued, and the final evaluation completed. |
| 2.22. | Exit Visual Acuity | Record the distance exit visual acuity, to the nearest letter, with the contact lenses (OD, OS, OU). |
| | | Note that the distance visual acuity must be at least 0.18 logMAR OU for the lenses to be dispensed and the participant must indicate that their vision is acceptable with the lenses. If the participant does not obtain an acceptable visual response (subjective or objective) remove the lenses, complete the slit-lamp exam and Final |
| | | Evaluation. |
| 2.23. | Dispensing Criteria | For the participant to continue in the study, they must meet all three of the following criteria: • Distance Binocular Visual acuity is 0.18 or better • The lens fit is acceptable OD and OS • Investigator approval. |
| | | If the Investigator does not approve the dispensing of the study lens, then the study is terminated for that participant. |
| 2.24. | Lenses | Subjects will be dispensed enough lenses to last them until their next visit. Additional "spare" |

| | | lenses may be dispensed to the subject based on |
|---|---|---|
| | | the Investigators discretion. |
| | | Subjects are permitted to use Refresh Plus® CL rewetting drops with the study lenses. Use of any |
| | | other artificial tears/lubricating eye drops is not |
| | | permitted with study CLs. |
| 2.25. | Patient Instructions | Instruct the Subject the following: |
| | | The lenses will be worn on a daily wear daily disposable basis. |
| | | <ul> <li>Enough lenses will be dispensed to the subject</li> </ul> |
| | | to wear for the required number of days until |
| | | their follow-up visit Additional "spare" |
| | | lenses may be dispensed to the subject based |
| | | on the Investigators discretion. |
| | | Instruct the subject to bring back all unworn |
| | | study lenses. If determined necessary by the |
| | | Investigator Refresh Plus® sterile non- |
| | | preserved rewetting drops may be dispensed to |
| | | be used as needed for dryness. |
| | | Subjects will be instructed to wear lenses for a minimum of 6 hours a day every day during. |
| | | minimum of 6 hours a day every day during the study. |
| | | <ul> <li>Subjects will be instructed to wear their</li> </ul> |
| | | glasses (if applicable) when not wearing the |
| | | study lenses. |
| | | A patient instruction booklet will be provided. |
| | | <b>Note:</b> In the event a lens is lost or damaged, if no |
| | | spare lenses are available, the subject will return |
| | | to the investigator site for replacement. As much |
| | | as reasonably possible, a damaged lens should be returned to the investigational site and then |
| | | returned to the Sponsor. If lens damage is |
| | | present, complete the Product Quality Complaint |
| | | Form. The lens will be stored in labeled vial with sterile saline and returned to the Sponsor. |
| 2.26. | Wearing Schedule | The test lenses will be worn on a daily wear, daily |
| | | disposable basis. |
| | | Note: Instruct the Neophytes / Lapsed wearer |
| | | subjects to follow this wear schedule for wearing |
| | | the study lenses: |
| | | Dispensing day: 6 hours of wear |

| | | Day 1: 6-8 hours of wear Day 2: 6-10 hours of wear Day 3: 6-12 hours of wear Day 4 and subsequent days: 6 to all waking hours of wear Note: For this protocol a day of wear is considered to be a minimum of 6 hours. When not wearing the study lenses the participant should be instructed to only wear their glasses (If applicable). For the follow-up visit instruct the participant they must have worn the lenses for at least 2 hours. |
|---|---|---|
| 2.27. | Follow-up | The participant will be scheduled to return for their follow-up appointment in 7±3 days. |

The Subjects must present to Visit 3 wearing the study contact lenses for at least 2 hours prior to the visit. If the subject has not worn the lenses for at least 2 hours the subject should be rescheduled.

| | Visit 3: Treatment 1 Follow-up 1 | |
|---|---|---|
| Ste<br>p | Procedure | Details |
| 3.1. | Adverse Events and<br>Concomitant<br>Medications<br>Review | Record any changes in concomitant medications and any adverse events that may have occurred since the last scheduled study visit. |
| 3.2. | Subject Reported<br>Ocular Symptoms | If the participant reports ocular symptoms with<br>their lenses, they will be recorded in the Subject<br>Reported Ocular Symptoms eCRF |
| 3.3. | Wear time and<br>Compliance | Subject's compliance with wearing the study CLs will be recorded. Record the hours/day and day/week the participant has worn the study lenses and CL wear time on the day of follow-up |
| 3.4. | Pupil size (Over the CLs) | Measure and record pupil size in photopic & scotopic lighting using Pupilometer over the contact lenses. Measure OD and OS at distance, intermediate(1m) and near (40cm). |
| 3.5. | Subjective<br>Acceptance | Record whether the subject's distance and near vision with the lenses is acceptable. |

| 2 | Visit 3: Treatment 1 Follow-up 1 | |
|---|---|---|
| Ste<br>p | Procedure | Details |
| 3.6. | Entrance Distance<br>VA (CLs) | Record distance and near (40cm) logMAR high contrast VA with the study CLs: OD, OS, OU to the nearest letter. |
| 3.7. | Over-refraction | Perform a distance over-refraction OD and OS using loose lenses over CLs under ambient room illumination. The distance over-refraction may also be refined under binocular conditions. Record the results. The results of the distance over-refraction may also be checked for the impact on near vision under monocular and/or binocular conditions. |
| 3.8. | Determination of<br>Lens Optimization | If the subject's vision is unacceptable for at least one distance or the Investigator determines that the visual acuity or over-refraction are not acceptable then a lens modification must be made. Up to two attempts at lens optimization are permitted if necessary, in order to achieve an acceptable distance and near binocular performance for the participant, and to enable them to wear the study lenses. Follow the fitting guide and the lens fitting steps 2.10 to 2.15 in Visit 2, allowing for adequate settling time between lens changes. (*Note: If a participant vision is unacceptable or requires a study lens power that is not available, during a modification, they will be discontinued from the study. Complete the slit-lamp and Final Evaluation). |
| 3.9. | Lens Fit<br>Assessment: | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). The participant should not proceed to wear the lenses if any of the following is observed: • presence of limbal exposure (appearance of clear cornea) in any gaze • presence of edge lift • presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up). If either lens is deemed unacceptable, the participant will be discontinued from the study. |

| C: | Visit 3: Treatment 1 Follow-up 1 | | |
|---|---|---|---|
| Ste<br>p | Procedure | Details | |
| | | Remove the lenses, perform a slit-lamp | 170 |
| | | evaluation, and complete the Final Evaluation | |
| | | form. | |
| 3.10. | Collection of | Collect unworn lenses returned by the subject | |
| | unworn lenses (if applicable) | when lens power has been optimized | |
| | | Note: If lens power was not changed allow the | |
| | | subject to use the unworn lenses dispensed at Visit | |
| | | 2 and dispense enough lenses of the same power | |
| | and of present to a contract to the contract of the contract o | to last the subject until their next visit. | |
| | Lens Removal | Remove and discard the lenses. | |
| 3.12. | Biomicroscopy | Non-dilated Slit Lamp Biomicroscopy will be | |
| | | performed. If the clearance of the fluorescein | |
| | | needs to be expedited, preservative-free rewetting | |
| 2 12 | Insertion of Study | drops or saline may be instilled. Dispense the participant new lenses that match | |
| 3.13. | Lenses | the original distance and ADD power of the | |
| | Lenses | lenses that were removed in Step 3.11 above. | |
| 3 14 | Post-Fit PRO | Subjects will complete the PRO (MRD) Contact | |
| Э.14. | (MRD) | Lens performance questionnaires. | |
| | Questionnaire | Ecos performance questionnanes. | |
| 3.15. | | Record Stereo-acuity using Near Stereo-Acuity | |
| | (40 cm) with CLs | test with CLs. | 2006 |
| 3.16. | Contrast Threshold | Record distance contrast threshold with CLs: OD, | |
| | (CLs) | OS and OU with the study contact lenses | |
| 3.17. | Pre-lens NITBUT | Measure and record NITBUT with Placido disc | |
| | | topographer projecting onto pre-lens tear film. OD, OS. | |
| 3.18. | Objective | Record objective accommodation using WAM | |
| | accommodation | 5500 refractometer for 4m, 1m, and 40cm targets | |
| | (CLs) | with the CLs. OD, OS. Record the average for | |
| | | each distance measurement OD, OS. | |
| 3.19. | | Measure the ocular aberrations using COAS, 2 | |
| | (over the CLs) | secs after blink, OD & OS @ distance target | |
| 2.00 | T1 (1 | Coma over the Contact lenses. | |
| 3.20. | 1 0 1 | Imaging for lens centration using Medmont | |
| 3.21. | centration) Exit Distance | Topographer, over CLs: OD, OS Record the distance visual acuity, to the nearest | |
| 3.41. | HCVA | letter, with the contact lenses (OD, OS, OU). | |
| | -10 111 | in the contact tenses (ob, oo, oo). | |
| | | Note that the distance visual acuity must be at | |
| | | least 0.18 logMAR OU for the lenses to be | |
| | | dispensed and the participant must indicate that | |

| | Visit 3: Treatment 1 Follow-up 1 | |
|---|---|---|
| Ste<br>p | Procedure | Details |
| | | their vision is acceptable with the lenses. If the participant does not obtain an acceptable visual response (subjective or objective) remove the lenses, complete the slit-lamp exam and Final Evaluation. |
| 3.22. | Dispensing Criteria | For the participant to continue in the study, they must meet all three of the following criteria: • Distance Binocular Visual acuity is 0.18 or better • The lens fit is acceptable OD and OS • Investigator approval. If the Investigator does not approve the dispensing |
| | | of the study lens, then the study is terminated for that participant. |
| 3.23. | Lenses | Subjects will be dispensed enough lenses to last them until their next visit. Additional "spare" lenses may be dispensed to the subject based on the Investigators discretion. Subjects are permitted to use Refresh Plus® CL rewetting drops with the study lenses. Use of any other artificial tears/lubricating eye drops is not permitted with study CLs. |
| 3.24. | Patient Instructions | <ul> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear daily disposable basis.</li> <li>Enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. Additional "spare" lenses may be dispensed to the subject based on the Investigators discretion. Instruct the subject to bring back all unworn study lenses.</li> <li>If determined necessary by the Investigator Refresh Plus ® sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day every day during the study.</li> </ul> |

| | Visit 3: Treatment 1 Follow-up 1 | |
|---|---|---|
| Ste<br>p | Procedure | Details |
| | | Subjects will be instructed to wear their glasses (if applicable) when not wearing the study lenses. Note: In the event a lens is lost or damaged, if no spare lenses are available, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with sterile saline and returned to the Sponsor. |
| 3.25. | Wearing Schedule | The test lenses will be worn on a daily wear, daily disposable basis. Note: For this protocol a day of wear is considered to be a minimum of 6 hours. When not wearing the study lenses the participant should be instructed to only wear their glasses (if applicable). For the follow-up visit instruct the participant they must have worn the lenses for at least 2 hours. |
| 3.26. | Follow-up | The participant will be scheduled to return for their follow-up (V4) appointment in 1 week ±3 days from visit #3. |

The Subjects must present to Visit 4 wearing the study contact lenses for at least 2 hours prior to the visit. If the subject has not worn the lenses for at least 2 hours the subject should be rescheduled.

| | Visit 4: Treatment 1 Follow-up 2 (2-week follow up) | |
|---|---|---|
| Step | Procedure | Details |
| 4.1. | Adverse Events and<br>Concomitant<br>Medications Review | Record any changes in concomitant medications and any adverse events that may have occurred since the last scheduled study visit. |
| 4.2. | Subject Reported<br>Ocular Symptoms | If the participant reports ocular symptoms with<br>their lenses, they will be recorded in the Subject<br>Reported Ocular Symptoms eCRF |
| 4.3. | Wear time and<br>Compliance | Subject's compliance with wearing the study CLs will be recorded. |

| | Visit 4: Treatment 1 Follow-up 2 (2-week follow up) | |
|---|---|---|
| Step | Procedure | Details |
| 4.4. | Follow-up PRO<br>(CLUE)<br>Questionnaire | Record the hours/day and day/ week the participant has worn the study lenses and CL wear time on the day of follow-up. Subjects will complete the PRO (CLUE) Contact Lens performance questionnaires. |
| 4.5. | Subjective<br>Acceptance | Record whether the subject's distance and near vision with the lenses is acceptable. Note: If the subject's distance and/or near vision is not acceptable with the study lenses the subject |
| 4.6. | Entrance LogMAR<br>HCVA Acuity | will be discontinued. Complete the Final Evaluation. Record the distance, intermediate (1M), and near logMAR visual acuity, to the nearest letter, with the contact lenses (OD, OS, OL) |
| 4.7. | Lens Fit Assessment | the contact lenses (OD, OS, OU). Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). The participant should not proceed to wear the lenses if any of the following is observed: • presence of limbal exposure (appearance of clear cornea) in any gaze • presence of edge lift • presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up). If either lens is deemed unacceptable, the participant will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form. |
| 4.8. | Stereo-acuity: near<br>(40 cm) CLs | Record Stereo-acuity using Near Stereo-Acuity test with CLs. |
| 4.9. | Contrast threshold<br>(CLs) | Record distance contrast threshold with CLs: OD, OS, and OU. |
| 4.10. | Pre-lens NITBUT | Measure and record NITBUT with Placido disc topographer projecting onto pre-lens tear film. OD, OS. |

| | Visit 4: Treatment 1 Follow-up 2 (2-week follow up) | |
|---|---|---|
| Step | Procedure | Details |
| 4.11. | Objective<br>accommodation<br>(CLs) | Record objective accommodation using WAM 5500 refractometer for 4m, 1m, and 40cm targets with the CLs. OD, OS. Record the average measurement for each distance OD, OS. |
| 4.12. | COAS<br>(over the CLs) | Measure the ocular aberrations using COAS 2 secs after blink, OD & OS @ distance target Coma over the Contact lenses. |
| 4.13. | Lens Removal | Remove and discard the lenses. |
| 4.14. | Biomicroscopy | Non-dilated Slit Lamp Biomicroscopy will be performed. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. |
| 4.15. | Continuance | Confirm the participant meets the criteria to continue. |
| 4.16. | Insertion of Study<br>Lenses | Dispense the participant new lenses that match the original distance and ADD power of the lenses that were removed in Step 4.13 above. Note: If the subject has unworn lenses from Visit 3 allow the subject to use the unworn lenses and dispense enough lenses of the same power to last the subject until their next visit. |
| 4.17. | Exit Distance HCVA | Record the distance visual acuity, to the nearest letter, with the contact lenses (OD, OS, OU). Note that the distance visual acuity must be at least 0.18 logMAR OU for the lenses to be dispensed and the participant must indicate that their vision is acceptable with the lenses. If the participant does not obtain an acceptable visual response (subjective or objective) remove the lenses, complete the slit-lamp exam and Final Evaluation. |
| 4.18. | Dispensing Criteria | For the participant to continue in the study, they must meet all three of the following criteria: • Distance Binocular Visual acuity is 0.18 or better • The lens fit is acceptable OD and OS • Investigator approval. |

| | Visit 4: Treatment 1 Follow-up 2 (2-week follow up) | |
|---|---|---|
| Step | Procedure | Details |
| | | If the Investigator does not approve the dispensing of the study lens, then the study is terminated for that participant. |
| 4.19. | Lenses | Subjects will be dispensed enough lenses & solutions to last them until their next visit. Additional "spare" lenses may be dispensed to the subject based on the Investigators discretion. Subjects are permitted to use Refresh Plus® CL rewetting drops with the study lenses. Use of any other artificial tears/lubricating eye drops is not permitted with study CLs. |
| 4.20. | Patient Instructions | <ul> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear daily disposable basis.</li> <li>Enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. Additional "spare" lenses may be dispensed to the subject based on the Investigators discretion. Instruct the subject to bring back all unworn study lenses.</li> <li>If determined necessary by the Investigator Refresh Plus® sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day every day during the study.</li> <li>Subjects will be instructed to wear their glasses (if applicable) when not wearing the study lenses.</li> <li>Note: In the event a lens is lost or damaged, if no spare lenses are available, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with</li> </ul> |

| | Visit 4: Treatment 1 Follow-up 2 (2-week follow up) | |
|---|---|---|
| Step | Procedure | Details |
| 4.21. | Wearing Schedule | The test lenses will be worn on a daily wear, daily disposable basis. Note: For this protocol a day of wear is considered to be a minimum of 6 hours. When not wearing the study lenses the participant should be instructed to only wear their glasses (if applicable). For the follow-up visit instruct the participant they must have worn the lenses for at least 2 hours. |
| 4.22. | Follow-up | The participant will be scheduled to return for their follow-up (V5) appointment in 4 weeks ±6 days from visit #4. |

The Subjects must present to Visit 5 wearing the study contact lenses for at least 2 hours prior to the visit. If the subject has not worn the lenses for at least 2 hours the subject should be rescheduled.

| | Visit 5: Treatment 1 Follow-up 3 (6-week follow up) | | |
|---|---|---|---|
| Ste | Procedure | Details | |
| p | | | |
| 5.1. | Adverse Events and | Record any changes in concomitant medications | 199 |
| | Concomitant | and any adverse events that may have occurred | |
| | Medications | since the last scheduled study visit. | |
| | Review | 52 | |
| 5.2. | Subject Reported | If the participant reports ocular symptoms with | |
| | Ocular Symptoms | their lenses, they will be recorded in the Subject | |
| | | Reported Ocular Symptoms eCRF | |
| 5.3. | Wear time and | Subject's compliance with wearing the study CLs | |
| | Compliance | will be recorded. | |
| | • | | |
| | | Record the hours/day and day/ week the | |
| | | participant has worn the study lenses and CL | |
| | | wear time on the day of follow-up. | |
| 5.4. | Follow-up PRO | Subjects will complete the PRO (CLUE) Contact | |
| | (CLUE) | Lens performance questionnaires. | |
| | Questionnaire | | |
| 5.5. | es un es | Record whether the subject's distance and near | |
| THE OWNER OF THE PARTY OF THE P | Subjective | vision with the lenses is acceptable. | |
| | Acceptance | | |
| | | L S | 8 |

| | Visit 5: Treatment 1 Follow-up 3 (6-week follow up) | |
|---|---|---|
| Ste<br>p | Procedure | Details |
| | | Note: If the subject's distance and/or near vision is not acceptable with the study lenses the subject will be discontinued. Complete the Final Evaluation. |
| 5.6. | Entrance LogMAR<br>HCVA Acuity | Record the distance intermediate (1M), and near logMAR visual acuity, to the nearest letter, with the contact lenses (OD, OS, OU). |
| 5.7. | Lens Fit<br>Assessment | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). The participant should not proceed to wear the lenses if any of the following is observed: • presence of limbal exposure (appearance of clear cornea) in any gaze • presence of edge lift • presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up). If either lens is deemed unacceptable, the participant will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation |
| 5.8. | Lens Removal | form. Remove and discard the lenses. |
| 5.9. | Biomicroscopy | Non-dilated Slit Lamp Biomicroscopy will be performed. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. |
| 5.10. | Continuance | Confirm the participant meets the criteria to continue. |
| 5.11. | Insertion of Study<br>Lenses | Dispense the participant new lenses that match the original distance and ADD power of the lenses that were removed in Step 5.8 above. Note: If the subject has unworn lenses from Visit 4 allow the subject to use the unworn lenses and dispense enough lenses of the same power to last the subject until their next visit. |
| 5.12. | Exit LogMAR<br>HCVA Acuity | Record the distance visual acuity, to the nearest letter, with the contact lenses (OD, OS, OU). |

| | Visit 5: Treatment 1 Follow-up 3 (6-week follow up) | |
|---|---|---|
| Ste | Procedure | Details |
| | | Note that the distance visual acuity must be at least 0.18 logMAR OU. for the lenses to be dispensed and the participant must indicate that their vision is acceptable with the lenses. If the participant does not obtain an acceptable visual response (subjective or objective) remove the lenses, complete the slit-lamp exam and Final Evaluation. |
| 5.13. | Dispensing Criteria | For the participant to continue in the study, they must meet all three of the following criteria: • Distance Binocular Visual acuity is 0.18 or better • The lens fit is acceptable OD and OS • Investigator approval. |
| | | If the Investigator does not approve the dispensing of the study lens, then the study is terminated for that participant. |
| 5.14. | Lenses / Solutions | Subjects will be dispensed enough lenses & solutions to last them until their next visit. Additional "spare" lenses may be dispensed to the subject based on the Investigators discretion. Subjects are permitted to use Refresh Plus® CL rewetting drops with the study lenses. Use of any other artificial tears/lubricating eye drops is not permitted with study CLs. |
| 5.15. | Patient Instructions | <ul> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear daily disposable basis.</li> <li>Enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. Additional "spare" lenses may be dispensed to the subject based on the Investigators discretion. Instruct the subject to bring back all unworn study lenses.</li> <li>If determined necessary by the Investigator Refresh Plus® sterile non-preserved rewetting drops may be dispensed to be used as needed</li> </ul> |

| | Visit 5: Treatment 1 Follow-up 3 (6-week follow up) | |
|---|---|---|
| Ste<br>p | Procedure | Details |
| | | <ul> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day every day during the study.</li> <li>Subjects will be instructed to wear their glasses (if applicable) when not wearing the study lenses.</li> </ul> |
| | | Note: In the event a lens is lost or damaged, if no spare lenses are available, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with sterile saline and returned to the Sponsor. |
| 5.16. | | The test lenses will be worn on a daily wear, daily disposable basis. Note: For this protocol a day of wear is considered to be a minimum of 6 hours. When not wearing the study lenses the participant should be instructed to only wear their glasses (if applicable). For the follow-up visit instruct the participant they must have worn the lenses for at least 2 hours. |
| 5.17. | Follow-up | The participant will be scheduled to return for their follow-up (V6) appointment in 6 weeks ±6 days from visit #5. |

The Subjects must present to Visit 6 wearing the study contact lenses for at least 2 hours prior to the visit. If the subject has not worn the lenses for at least 2 hours the subject should be rescheduled.

| | Visit 6: Treatment 1 Follow-up 4 (12-week follow up) | |
|---|---|---|
| Step | Procedure | Details |
| 6.1. | Adverse Events and<br>Concomitant<br>Medications<br>Review | Record any changes in concomitant medications and any adverse events that may have occurred since the last scheduled study visit. |

| | Visit 6: Treatment 1 Follow-up 4 (12-week follow up) | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 6.2. | Subject Reported<br>Ocular Symptoms | If the participant reports ocular symptoms with<br>their lenses, they will be recorded in the Subject<br>Reported Ocular Symptoms eCRF | |
| 6.3. | Wear time and<br>Compliance | Subject's compliance with wearing the study CLs will be recorded. Record the hours/day and day/ week the participant has worn the study lenses and CL wear time on the day of follow-up. | |
| 6.4. | Collection of unworn lenses | Collect unworn lenses returned by the participant. | * |
| 6.5. | Follow-up PRO<br>(CLUE & MRD)<br>Questionniares | Subjects will complete PRO (CLUE and MRD) Contact Lens performance questionnaires. | |
| 6.6. | Subjective<br>Acceptance | Record whether the subject's distance and near vision with the lenses is acceptable. | |
| 6.7. | Entrance LogMAR<br>HCVA Acuity | Record the distance, intermediate (1M), and near logMAR visual acuity, to the nearest letter, with the contact lenses (OD, OS, OU). | |
| 6.8. | Lens Fit Assessment | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). The participant should not proceed to wear the lenses if any of the following is observed: • presence of limbal exposure (appearance of clear cornea) in any gaze • presence of edge lift • presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up). If either lens is deemed unacceptable, the participant will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form. | |
| 6.9. | Stereo-acuity: near<br>(40 cm) CLs | Record Stereo-acuity using Near Stereo-Acuity test with CLs. | |
| 6.10. | Contrast threshold (CLs) | Record distance contrast threshold with CLs: OD, OS, and OU. | |
| 6.11. | Objective accommodation | Record objective accommodation using WAM 5500 refractometer for 4m, 1m, and 40cm targets | |

| | Visit 6: Treatment 1 Follow-up 4 (12-week follow up) | |
|---|---|---|
| Step | Procedure | Details |
| | (CLs) | with the CLs. OD, OS. Record the average measurement for each distance OD, OS. |
| 6.12. | COAS<br>(over the CLs) | Measure the ocular aberrations using COAS 2 secs after blink, OD & OS @ distance target Coma over the Contact lenses. |
| 6.13. | Lens Removal | Remove and discard the lenses. |
| 6.14. | Biomicroscopy | Non-dilated Slit Lamp Biomicroscopy will be performed. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. |

# **Final Evaluation**

| | Final Evaluation | |
|---|---|---|
| Step | Procedure | Details |
| F.1 | Post-fit Interview Study CL Performance Occupation Hobbies, Visual Demands, Success Criteria, Reasons for Success/Failure | Questions regarding the study CL performance for the participant's: occupation and hobbies Visual demands, eg laptop, shift work, night driving etc. Success criteria with the study CL Factors affecting success/failure with the study CL |
| F.2 | Investigator<br>Recommendation | Investigator recommendation, if applicable (study CLs suitable/not suitable to prescribe, plus investigator reasons where not suitable is indicated) Proceed with final evaluation |
| F.3 | Distance Subjective<br>Sphero-cylindrical<br>Refraction | Perform an optimal monocular/binocular distance<br>best sphero-cylindrical refraction and record the<br>visual acuity (OD, OS, OU) to the nearest letter<br>(this is referred to as the best corrected visual<br>acuity, BCVA). |
| F.4 | Subject Disposition | Indicate the participant completed the study successfully or not. For subjects who discontinue, indicate the reason. |
| F.5 | PRO (CLUE &<br>MRD)<br>Questionnaires | Subjects will complete the PRO (CLUE and MRD) contact lens performance questionnaires. |

| | Final Evaluation | |
|---|---|---|
| Step | Procedure | Details |
| | (Discontinued | |
| | Subjects Only) | |
| F.6 | Biomicroscopy | Non-dilated Slit Lamp Biomicroscopy will be |
| | (Discontinued | performed. |
| | Subjects if not | If the clearance of the fluorescein needs to be |
| | completed during | expedited, preservative-free rewetting drops or |
| | the visit) | saline may be instilled. |

### 7.3. Unscheduled Visits

If, during the investigation, a participant requires an unscheduled visit to the clinical site, the following information will be collected at a minimum:

- Chief complaint prompting the visit. If the reason is an adverse event, the applicable eCRF for the adverse event must be completed and participant record completed as appropriate
- Date and time of the visit and all procedures completed at the unscheduled visit
- Review of adverse event and concomitant medications
- Documentation of any test article dispensed or collected from the participant, if applicable
- Slit lamp findings (using the Slit Lamp Classification Scale)

If the Investigator withdraws a participant from the study, the final study visit case report forms must be completed indicating the reason(s) why the participant was withdrawn. The participant record must be completed documenting the date and primary reason for withdrawal and the study CRA notified.

Any ocular and non-ocular Adverse Events that are ongoing at the time of the study visit will be followed by the Investigator, within licensure, until they have resolved, returned to pretreatment status, stabilized, or been satisfactorily explained. If further treatment i.e., beyond licensure is required, the participant will be referred to the appropriate health care provider.

The following information may be collected during an unscheduled visit as required.

| | Unscheduled Visit | | |
|---|---|---|---|
| Step | Procedure | Details | 10 m |
| U.1 | Chief Complaints | Record the participant's chief complaints for reasons for the unscheduled visit. | 200 |
| U.2 | Adverse Events and<br>Concomitant<br>Medications Review | Review any changes to the participant's medical history or concomitant medications from the previous study visit. Record any changes, and any adverse events. | |

| | | Unscheduled Visit |
|---|---|---|
| Step | Procedure | Details Details |
| U.3 | Subject Reported<br>Ocular Symptoms | If the participant reports ocular symptoms with their lenses, they will be recorded in the |
| U.4 | Entrance logMAR<br>HCVA | Record the entrance distance visual acuity (OD, OS and OU) to the nearest letter. |
| U.5 | Subjective Sphero-<br>cylindrical<br>Refraction | Perform bare-eye subjective spherocylindrical refraction with a phoropter (adopt the maximum plus to maximum visual acuity (MPMVA) approach and use the duo-chrome test for binocular balancing) and record the best corrected distance visual acuity to the nearest letter (OD, OS, and OU). |
| U.6 | Biomicroscopy | Non-dilated Slit Lamp Biomicroscopy will be performed. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. |
| U.7 | Lens Fit Assessment | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). The participant should not proceed to wear the lenses if any of the following is observed: • presence of limbal exposure (appearance of clear cornea) in any gaze • presence of edge lift • presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up). If either lens is deemed unacceptable, the participant will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form. |
| U.8 | Exit logMAR HCVA | Record the participant's exit distance visual acuity (OD, OS, and OU) to the nearest letter. |
| U.9 | Dispensing Criteria | For the participant to continue in the study, they must meet all three of the following criteria: • Distance Binocular Visual acuity is 0.18 or better • The lens fit is acceptable OD and OS • Investigator approval. |

| | Unscheduled Visit | |
|---|---|---|
| Step | Procedure | Details |
| U.10 | Dispensing of<br>Lenses / Solutions (if<br>applicable) | If the Investigator does not approve the dispensing of the study lens, then the study is terminated for that participant. Subjects will be dispensed enough lenses & solutions to last them until their next visit. Subjects are permitted to use Refresh Plus® |
| | | their habitual CL rewetting drops with the study lenses. Use of any other artificial tears/lubricating eye drops is not permitted with study CLs. |
| U.11 | Patient Instructions (if applicable) | <ul> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear daily disposable basis.</li> <li>Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. No additional lenses will be dispensed.</li> <li>Instruct the subject to bring back all unworn study lenses.</li> <li>If determined necessary by the Investigator Refresh Plus® sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day every day during the study.</li> <li>Subjects will be instructed to wear their glasses (if applicable) when not wearing the study lenses.</li> <li>A patient instruction booklet will be provided.</li> <li>Note: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present,</li> </ul> |

| Unscheduled Visit | | |
|---|---|---|
| Step | Procedure | Details |
| | | Form. The lens will be stored in labeled vial with sterile saline and returned to the Sponsor. |
| U.12 | Wear Schedule for | The test lenses will be worn on a daily wear, |
| | Neophytes / Lapsed | daily disposable basis. |
| | Wearers | |
| | | Note: Instruct the Neophytes / Lapsed |
| | | wearer subjects to follow this wear schedule |
| | | for wearing the study lenses: |
| | | Dispensing day: 6 hours of wear |
| | | Day 1: 6-8 hours of wear |
| | | Day 2: 6-10 hours of wear |
| | | Day 3: 6-12 hours of wear |
| | | Day 4 and subsequent days: 6 to all waking |
| | | hours of wear |
| | | Note: For this protocol a day of wear is |
| | | considered to be a minimum of 6 hours. When |
| | | not wearing the study lenses the participant |
| | | should be instructed to only wear their |
| | | glasses (If applicable). For the follow-up |
| | | visit instruct the participant they must have |
| | | worn the lenses for at least 2 hours. |

## 7.4. Laboratory Procedures

Not applicable. There will be No Laboratory Procedures in this study.

## 8. SUBJECTS COMPLETION/WITHDRAWAL

## 8.1. Completion Criteria

Subjects are considered to have completed the study if they:

- provided informed consent
- they are eligible
- they have completed all 6 study visits (V1-V6) through the final visit
- have not withdrawn/discontinued from the study for any reason described in Section 8.2

# 8.2. Withdrawal/Discontinuation from the Study

A participant will be withdrawn from the study for any of the following reasons:

- Participant death during the study period
- Participant withdrawal of consent

- Participant not compliant to protocol (not compliant with or not able to follow study procedures, or study procedures/interviews /assessments could not be conducted)
- Participant lost to follow-up
- Participant no longer meets eligibility criteria (e.g. the participant becomes pregnant)
- Participant develops significant or serious adverse event during the study visit (e.g. a heart attack)
- Subjects presenting with a Corneal Infiltrative Event (CIE), or an eye infection
- Subject develops significant or serious adverse events causing discontinuation of study lens wear (missing more than half of the required days of lens wear in-between visits will lead to discontinuation, e.g. wearing the lens for only 1 day instead of the minimum of 4 days between visits 2 and 3)
- Investigator's clinical judgment regarding the participant safety reasons (that it is in the best interest of the participant to stop the study visit)
- Participant missed two consecutive study visits
- Participant not compliant with study lens wear schedule
- Participant not successfully dispensed due to lack of efficacy and safety including poor vision, poor comfort or unacceptable fit

For discontinued Subjects, the Investigator will:

- not complete the scheduled visit procedures
- Complete the Final Evaluation, indicating the reason that the participant was discontinued from the study
- Record the spherocylindrical refraction with best corrected distance visual acuity if applicable (i.e. if this was already measured during the same day) otherwise perform a spherocylindrical refraction and record the exit distance visual acuity.
- Collect used test article(s) (worn or brought to the visit) from the participant and discard them, unless otherwise stated in Section 7.2
- Collect all unused test article(s) from the participant

An additional participant may be enrolled if a participant discontinues from the study prematurely.

In cases where a participant is lost to follow-up, every possible effort must be made to contact the participant and determine the reason for discontinuation/withdrawal. The measures taken to follow up must be documented including two written attempts and a certified letter (or equivalent) as the final attempt.

### 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION

Concomitant medications will be documented during screening and updated during the study. Disallowed medications for this study include: Any topical ocular medications except lubricating eye drops.

Concomitant therapies that are disallowed include: A change within the previous 3 months to the dosage of a systemic medication known to affect prescription or ocular surface or tear film (eg. steroids).

#### 10. DEVIATIONS FROM THE PROTOCOL

Investigator will notify study sponsor upon identification of a protocol deviation. Major protocol deviations must be reported to the sponsor within 24 hours after discovery of the protocol deviation. The Investigator will report deviations per IRB/IEC requirements. All deviations will be tracked, and corrective actions implemented as appropriate.

If it becomes necessary for the Investigator to implement a deviation in order to eliminate an immediate hazard to the trial participant, the Investigator may implement the deviation immediately without notification to the sponsor. Within 24 hours after the implemented deviation, the Investigator must notify and provide the rationale to the Sponsor and, as required, the IEC/IRB.

#### 11. STUDY TERMINATION

The occurrence of one or more Unanticipated Serious Adverse Device Effect (USADE), or any SAE where the relationship to study agent cannot be ruled out, may result in stopping further dispensing of test article. In the event of a USADE or SAE, the Sponsor may unmask (if applicable) the treatment regimen for the participant(s) and will discuss this with the Investigator before any further Subjects are enrolled.

The Sponsor will determine when a study will be stopped. The Principal Investigator always has the discretion to initiate stopping the study based on patient safety or if information indicates the study's results are compromised.

JJVC reserves the right to terminate the study at any time for any reason. Additionally, the IEC/IRB reserves the right to terminate the study if an unreasonable risk is determined. The study can be terminated by the Principal Investigator at the individual clinical site due to specific clinical observations, if in their opinion, after a discussion with JJVC, it is determined that it would be unwise to continue at the clinical site.

JJVC (and the IEC/IRB and DMC, if applicable) will evaluate all adverse events. If it is determined that an adverse event presents an unreasonable risk, the investigation, or that part of the investigation presenting the risk, will be terminated, as soon as possible.

Should the study be terminated (either prematurely or as scheduled), the Investigator will notify the IEC/IRB and Regulatory Authority as required by local regulatory requirements.

# 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS

A Product Quality Complaint (PQC) refers to any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness or performance of test articles after they have been released for clinical trial use.

Potential complaints may come from a variety of sources including but not limited to Subjects, clinical research associates (CRA), clinical operations managers (COM), medical monitors, and site personnel, etc. The following are not considered product quality complaints:

- Subject satisfaction inquiries reported via "Subjective Questionnaires" and "Patient Reported Outcomes (PRO)"
- Clinical test articles that are stored improperly or damaged after receipt at the investigational site
- Lens replacements that occur due to drops/fall-outs
- Damage deemed by clinicians or clinical staff to be caused by handling by the user, and not indicative of a quality deficiency (i.e. tears, rips, etc.), only in situations where there is no deficiency alleged by the participant

Within 24 hours of site personnel becoming aware that a PQC has occurred, the PQC must be recorded in the EDC system, which will trigger an automatic email notification to the appropriate COM/CRA and Clinical QA representative. In cases where the EDC system in use is not configured to send automatic notifications or when an EDC system is not used, the COM/CRA is responsible for notifying Clinical QA upon discovery that a PQC has occurred.

Upon receipt of the EDC notification, the COM/CRA will contact the study site to collect additional information which will include:

- Date the complaint was received/recorded in the EDC System (Date of Sponsor Awareness)
- Who received the complaint
- Study number
- Clinical site information (contact name, site ID, telephone number)
- Lot number(s)
- Unique Subject Identifier(s)
- Indication of who first observed complaint (site personnel or participant)
- OD/OS indication, along with whether the lens was inserted
- Any related AE number if applicable
- Detailed complaint description (scheduled/unscheduled visit, wear time, symptoms, resolution of symptoms, etc.)
- Eye Care Provider objective (slit lamp) findings if applicable
- Confirmation of product availability for return (and tracking information, if available), or rationale if product is not available for return

Once a complaint is received, it will be assessed by the COM, CRA, or trained site personnel to determine if it is an Adverse Event/Serious Adverse Event (AE/SAE). If the complaint results in an AE/SAE, the COM/CRA, or trained site personnel will follow Section 13 of this protocol. If the AE/SAE was potentially the result of a product quality related deficiency, these procedures also applies and will be executed in parallel.

In some cases, a PQC form may be generated in EDC by the site in error. In this event, the PQC forms will be marked "Intentionally Left Blank" or "ILB". Justification for ILB must be documented.

#### 13. ADVERSE EVENTS

### 13.1. Definitions and Classifications

**Adverse Event (AE)** – An AE is "any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in Subjects, users or other persons, whether or not related to the investigational medical device.

*Note 1* to entry: This definition includes events related to the investigational medical device or the comparator.

*Note 2* to entry: This definition includes events related to the procedures involved.

*Note 3* to entry: For users or other persons, this definition is restricted to events related to investigational medical devices."<sup>1</sup>

An AE includes any condition (including a pre-existing condition) that:

- 1. Was not present prior to the study, but appeared or reappeared following initiation of the study
- 2. Was present prior to the study but worsened during the study. This would include any condition resulting from concomitant illnesses, reactions to concomitant medications, or progression of disease states
- 3. Pregnancy must be documented as an adverse event and must be reported to the clinical monitor and to the Sponsor immediately upon learning of the event

**Serious Adverse Event (SAE)** – An SAE is any untoward medical occurrence that:

- Results in death
- Is life threatening
- Requires in-patient hospitalization or prolongation of existing hospitalization

Results in persistent or significant disability/incapacity (e.g., a sight threatening event, a significant persistent or permanent change, impairment, damage, or disruption to the participant's body)

- Is a congenital anomaly/birth defect
- Requires intervention to prevent permanent damage (the use of the test article resulting in a condition which requires medical or surgical intervention to preclude permanent impairment of the body structure or a body function). Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered an SAE when, based upon appropriate medical judgment, they may jeopardize the patient or participant and may require medical or surgical intervention to prevent one of the outcomes listed in the above definition

Diagnoses and conditions that are considered Ocular Serious Adverse Events include, but not limited to:

- Microbial Keratitis (MK)
- Iritis (including cells in the anterior chamber)
- Permanent decrease in best spectacle corrected visual acuity (BSCVA) equivalent to 2 acuity lines or greater
- Central Corneal Opacity
- Central Corneal Neovascularization

- Uveitis
- Endophthalmitis
- Hypopyon
- Hyphemia
- Penetration of Bowman's Membrane
- Persistent Epithelial Defect
- Limbal cell Damage leading to Conjunctivalization

**Significant Adverse Events** – Those events that are usually symptomatic and warrant discontinuation (temporary or permanent) of the test article (excluding Serious Adverse Events).

Diagnoses and conditions that are considered Ocular Significant Adverse Events include, but not limited to the following:

- Contact Lens Induced Peripheral Ulcer (CLPU)
- Significant Infiltrative Events (SIE)
- Superior Epithelial Arcuate Lesions (SEALs)
- Any Temporary Loss of >2 Lines of BSCVA
- Other grade 3 or higher corneal findings, such as abrasions or edema
- Non-contact lens related corneal events e.g. Epidemic Keratoconjunctivitis (EKC)
- Asymptomatic Corneal Scar
- Any corneal event which necessitates temporary lens discontinuation >2 weeks

**Non-Significant Adverse Events** — Those conditions that are usually asymptomatic and usually do not warrant discontinuation (temporary or permanent) of the test article. However, the Investigator may choose to treat as a precautionary measure.

Diagnoses and conditions that are considered Ocular Non-Significant Adverse Events include, but not limited to the following:

- Non-significant Infiltrative Event (NSIE)
- Contact Lens Papillary Conjunctivitis (CLPC)
- Superficial Punctate Keratitis (SPK)
- Conjunctivitis: Bacterial, Viral, Allergic
- Blepharitis
- Meibomianitis
- Contact Dermatitis
- Localized Allergic Reactions
- Any corneal event not explicitly defined as serious or significant adverse event, which necessitates temporary lens discontinuation < 2 weeks

**Adverse Device Effect (ADE)** – An ADE is an "adverse event related to the use of an investigational medical device.

*Note 1* to entry: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device.

*Note 2* to entry: This definition includes any event resulting from use error or from intentional misuse of the investigational medical device."

Unanticipated Adverse Device Effect (UADE) – Any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, the test article, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan, Investigator's Brochure or protocol, or any other unanticipated serious problem associated with the test article that relates to the rights, safety and welfare of Subjects.

### 13.2. Assessing Adverse Events

In conjunction with the medical monitor, the Investigator will evaluate adverse events to ensure the events are categorized correctly. Elements of categorization will include:

- Seriousness/Classifications (see definition in Section 13.1)
- Causality or Relatedness i.e. the relationship between the test article, study treatment or study procedures and the adverse event (not related; unlikely related; possibly related; related see definition in Section 13.2.1)
- Adverse Event Severity Adverse event severity is used to assess the degree of intensity of the adverse event (mild; moderate; severe for all events - see definition in Section 13.2.2)
- Outcome not recovered or not resolved; recovering or resolving; recovered or resolved with sequelae; recovered or resolved; death related to adverse event; unknown
- Actions Taken none; temporarily discontinued; permanently discontinued; other

### 13.2.1. Causality Assessment

**Causality Assessment** – A determination of the relationship between an adverse event and the test article. The test article relationship for each adverse event should be determined by the investigator using these explanations:

- Not Related- An adverse event that is not related to the use of the test article, study treatment or study procedures
- Unlikely Related An adverse event for which an alternative explanation is more likely, e.g. concomitant treatment, concomitant disease(s), or the relationship of time suggests that a causal relationship is not likely
- Possibly Related An adverse event that might be due to the use of the test article, or to the study treatment or study procedures. An alternative explanation, e.g. concomitant treatment, concomitant disease(s), is inconclusive. The relationship in time is reasonable. Therefore, the causal relationship cannot be excluded
- Related An adverse event that is listed as a possible adverse effect (device) or adverse reaction (drug) and cannot be reasonably explained by an alternative explanation, e.g. concomitant treatment of concomitant disease(s). The relationship in time is very suggestive, e.g. it is confirmed by de-challenge and re-challenge

### 13.2.2. Severity Assessment

**Severity Assessment** – A qualitative assessment of the degree of intensity of an adverse event as determined by the Investigator or reported to him/her by the participant. The assessment of

severity is made irrespective of test article, study treatment or study procedure relationship or seriousness of the event and should be evaluated according to the following scale:

- Mild Event is noticeable to the participant, but is easily tolerated and does not interfere with the participant's daily activities
- Moderate Event is bothersome, possible requiring additional therapy, and may interfere with the participant's daily activities
- Severe Event is intolerable, necessitates additional therapy or alteration of therapy and interferes with the participant's daily activities

# 13.3. Documentation and Follow-Up of Adverse Events

The recording and documenting of adverse events (ocular and non-ocular) begins when the Subjects are exposed to the test article, study treatment or study procedure. Adverse events reported before the use of test article, start of study treatment, or study procedures will be recorded as medical history. However, if the condition deteriorates at any time during the study it will be recorded and reported as an AE. Untoward medical events reported after the participant's exit from the study will be recorded as adverse events at the discretion of the Investigator.

Upon finding an adverse event, the Principal Investigator will document the condition in the participant record and in the eCRFs. He/she will complete the Adverse Event /eCRF.

Complete descriptions of all adverse events must be available in the participant record. All Adverse Events including local and systemic reactions not meeting the criteria for "serious adverse events" shall be captured on the appropriate case report form or electronic data system. All adverse events occurring while the participant is enrolled in the study must be documented appropriately regardless of relationship.

It is the Investigator's responsibility to maintain documentation of each reported adverse event. All adverse events will be followed in accordance with applicable licensing requirements. Such documentation will include the following:

- Adverse event (diagnosis not symptom)
- Drawings or photographs (where appropriate) that detail the finding (e.g., size, location, and depth, etc.)
- Date the clinical site was notified
- Date and time of onset
- Date and time of resolution
- Adverse event classification, severity, and relationship to test articles, as applicable
- Treatment regimen instituted, including concomitant medications prescribed, in accordance with applicable licensing requirements
- Any referral to another health care provider if needed
- Outcome, ocular damage (if any)
- Likely etiology
- Best corrected visual acuity at the discovery of the event and upon conclusion of the event

In addition, if an infiltrate(s) is present, he/she will complete the Corneal Infiltrate Assessment eCRF. Where necessary, a culture of the corneal lesion will be collected to determine if the infection is microbial in nature. If cultures are collected, the date of culture collection and laboratory utilized will be recorded.

Changes in the severity of an AE shall be documented to allow an assessment of the duration of the event at each level of intensity to be performed. Adverse events characterized as intermittent require documentation of the onset and duration of each episode. Changes in the assessment of relationship to the Test Article shall also be clearly documented.

Subjects who present with an adverse event shall be followed by the Investigator, within licensure, until all signs and symptoms have returned to pre-treatment status, stabilized, or been satisfactorily resolved. If further treatment beyond licensure is required, the patient will be referred to the appropriate health care provider. The Investigator will use his/her clinical judgment as to whether a participant reporting with an adverse event will continue in the study. If a participant is discontinued from the study, it will be the responsibility of the Investigator to record the reason for discontinuation. The Investigator will also document the adverse event appropriately and complete the Adverse Event eCRF. Any Subjects with ongoing adverse events related to the test article, study treatment or study procedures, as of the final study visit date, should be followed to resolution of the adverse event or until referral to an appropriate health care provider, as recommended by the Investigator. Non-ocular adverse events that are not related to the test article, study treatment, or study procedures may be recorded as "ongoing" without further follow-up.

### 13.4. Reporting Adverse Events

The Investigator will notify the Sponsor of an adverse event by e-mail, facsimile, or telephone as soon as possible and no later than 24 hours from discovery for any serious /significant adverse events, and 2 days from discovery for any non-significant adverse event. In addition, a written report will be submitted by the Principal Investigator to the IEC/IRB according to their requirements (Section 13.4.2). The report will comment whether the adverse event was considered to be related to the test article, study treatment or study procedures.

### 13.4.1. Reporting Adverse Events to Sponsor

### **Serious/Significant Adverse Events**

The Investigator will inform the sponsor of all serious/significant adverse events occurring during the study period as soon as possible by e-mail, fax, or telephone, but no later than 24 hours following discovery of the event. The Investigator is obligated to pursue and obtain information requested by the Sponsor in addition to that information reported on the eCRF. All Subjects experiencing a serious/significant adverse event must be followed up and all outcomes must be reported.

When medically necessary, the Investigator may break the randomization code (if applicable) to determine the identity of the treatment that the participant received. The Sponsor and study monitor should be notified prior to unmasking (if applicable) the test articles.

In the event of a serious/significant adverse event, the Investigator must:
- Notify the Sponsor immediately
- Obtain and maintain in the participant's records all pertinent medical information and medical judgment for colleagues who assisted in the treatment and follow-up of the participant
- Provide the Sponsor with a complete case history which includes a statement as to whether the event was or was not related to the use of the test article
- Notify the IEC/IRB as required by the IEC/IRB reporting procedure according to national regulations

# **Unanticipated (Serious) Adverse Device Effect (UADE)**

In the event of an Unanticipated (Serious) Adverse Device Effect (UADE), the Investigator will submit a report of the UADE to the Sponsor and IEC/IRB as soon as possible, but no later than 24 hours after the Investigator first learns of the effect. This report is in addition to the immediate notification mentioned above.

The Sponsor must conduct an evaluation of the UADE and must report the results of the evaluation to FDA, the IEC/IRB and participating Investigators within 10 working days after the Sponsor first receives notification of the effect.

#### **Non-Serious Adverse Events**

All non-serious adverse events, including non-serious adverse device effects, will be reported to the sponsor by the Investigator no later than 2 days from discovery.

# 13.4.2. Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities

Adverse events that meet the IEC/IRB requirements for reporting must be reported within the IEC/IRB's written guidelines. Each clinical site will refer to and follow any guidelines set forth by their Approving IEC/IRB. Each clinical site will refer to and follow any guidelines set forth by their local governing Health Authorities.

The Sponsor will report applicable Adverse Events to the local health authorities according the written guidelines, including reporting timelines.

## 13.4.3. Event of Special Interest

Not applicable - No events of special interest are expected for this study.

## 13.5. Reporting of Pregnancy

Subjects reporting pregnancy (by self-report) during the study screening section of this study will be discontinued as a screen failure. Subjects reporting pregnancy (by self-report) during the study will be discontinued after the event is recorded as an Adverse Event. Once discontinued, pregnant Subjects and their fetuses will not be monitored for study related purposes. Pregnant Subjects are not discontinued from contact lens or solution related studies for safety concerns, but due to general concerns relating to pregnancy and contact lens use. Specifically, pregnant women are discontinued due to fluctuations in refractive error and/or visual acuity that occur secondary to systemic hormonal changes, and not due to unforeseen health risks to the mother or fetus.


#### 14. STATISTICAL METHODS

## 14.1. General Considerations

Statistical Analysis will be undertaken by the sponsor. A general description of the statistical methods to be implemented in this clinical trial is outlined below.

All data summaries and statistical analyses will be performed using the SAS software Version 9.4 or higher (SAS Institute, Cary, NC). Throughout the analysis of data, the results for each subject/eye will be used when available for summarization and statistical analysis. Unscheduled visits will be summarized separately and will be excluded from the statistical analysis.

Summary tables (descriptive statistics and/or frequency tables) will be provided for all baseline variables, efficacy variables and safety variables as appropriate. Continuous variables will be summarized with descriptive statistics (n, mean, standard deviation [SD], median, minimum and maximum). Frequency count and percentage of subjects or eyes within each category will be provided for categorical data.

# 14.2. Sample Size Justification

This is an exploratory study to generate initial data for assessing a computational vision model. As such, the sample size was not determined based on any power analysis with regard to the primary endpoint. The collected data will be used to design future studies, if necessary.

The planned sample size (75 to enroll and 50 to complete) was selected to enroll different categories of myopic presbyopes including previous MF CL wearers, Single vision CL wearers and Subjects who are neophyte to CL wear. Efforts will be made to enroll subjects in all three categories without specific targets to be achieved.

All analysis will be conducted on the per-protocol population defined in section 14.3.

# 14.3. Analysis Populations

#### **Safety Population:**

All Subjects who were administered any test article excluding Subjects who drop out prior to administering any test article. At least one observation should be recorded.

## **Per-Protocol Population:**

All Subjects who have successfully completed all visits and did not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock (Per-Protocol Population). Justification of excluding Subjects with protocol deviations in the per-protocol population set will be documented in a memo to file.

## **Intent-to-Treat (ITT) Population:**

All Subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol. At least one observation should be recorded.

## 14.4. Level of Statistical Significance

All planned analysis for this study will be conducted with an overall type I error rate of 5%.

## 14.5. Primary Analysis

## Likelihood to be a successful lens wearer vs. Quest questionnaire classification

The successful lens wear will be converted to a binary response the same as in the previous analysis. The proportion of response ("1") will be analyzed using a generalized linear mixed model with a binary distribution and logit link function for all questions. Each model will include the experimental design factors: Quest questionnaire classification as the fixed effect; and subject as the random effect. Other baseline characteristics known to be important such as age, sex, and/or add power will be included as fixed covariates when appropriate.

The proportion of successful lens wear for the subjects classified as being "discontented and driven" will be calculated with 95% CI for least square mean. If the lower limit of the CI is greater than 75%, the statistical superiority will be concluded.

## 14.6. Secondary Analysis

## Likelihood to be a successful lens wearer vs. physical ocular related measurements

The secondary analysis will be conducted using the same method as descried in Section 14.5 regarding CLUE vision score at baseline. In the model the CLUE vision score at baseline will be replaced by the secondary endpoints (defined in Section 2.2) one at a time to determine the significance level of each physical ocular related measurement. If the measurement is taken by eye, average value of the left and right eye will be used.

Kenward and Roger<sup>6</sup> method will be used for the calculation of the denominator of degrees of freedom.

## 14.7. Other Exploratory Analyses

Not Applicable.

## 14.8. Interim Analysis

Not applicable.

## 14.9. Procedure for Handling Missing Data and Drop-Outs

Missing or spurious values will not be imputed. The count of missing values will be included in the summary tables and listings.

Subject dropout is expected to be one of the main reasons of missing data in this clinical trial. Past clinical trials don't provide the evidence that participant dropout is systematic or not-at-random. To evaluate the impact of missing data, sensitivity analysis will be conducted using multiple imputation methods if the proportion of participant dropout is greater than the 15%. The SAS/STAT procedures PROC MI and PROC MIANALYZE will be utilized with a parametric regression method used to make at least 5 imputations.

## 14.10. Procedure for Reporting Deviations from Statistical Plan

The analysis will be conducted according to that specified in above sections. There are no known reasons for which it is planned to deviate from these analysis methods. If for any reason a change is made, the change will be documented in the study report along with a justification for the change.

#### 15. DATA HANDLING AND RECORD KEEPING/ARCHIVING

## 15.1. Electronic Case Report Form/Data Collection

The data for this study will be captured on electronic case report forms (eCRFs) using the Bioclinica EDC system. An authorized data originator will enter study data into the eCRFs using the EDC system. Data collected on equipment that is not captured in EDC will be formatted to the specification of the JJVC database manager and sent to JJVC for analysis. Data generated from interviews will be saved as audio files and any subsequent collation and tabulation of the interview notes will be organized in both Word and Excel files.

Where applicable, data print-outs from instruments will be marked with study and participant identifiers and retained in the participant record. If the print-out ink/paper are not stable, they will be photocopied, and the photocopy will also be retained in the participant record.

External Date Sources for this study include: Not Applicable

The clinical data will be recorded on dedicated eCRFs specifically designed to match the study procedures for each visit. Once completed, the eCRFs will be reviewed for accuracy and completeness and signed by the Investigator. The sponsor or sponsor's representatives will be authorized to gain access to the participant recordation for the purposes of monitoring and auditing the study.

Edit checks, electronic queries, and audit trails are built into the system to ensure accurate and complete data collection. Data will be transmitted from the clinical site to a secure central database as forms are completed or updated, ensuring information accuracy, security, and confidentiality. After the final database lock, the Investigator will be provided with Individual Patient Profiles (IPP) including the full audit trail on electronic media in PDF format for all of the study data. The IPP must be retained in the study files as a certified copy of the source data for the study.

The content and structure of the eCRFs are compliant with ISO14155:2011.<sup>1</sup>

## 15.2. Subject Record

At a minimum, participant record should be available for the following:

- participant identification
- eligibility
- study identification
- study discussion
- provision of and date of informed consent
- visit dates
- results of safety and efficacy parameters as required by the protocol
- a record of all adverse events
- follow-up of adverse events
- medical history and concomitant medication
- test article receipt/dispensing/return records
- date of study completion
- reason for early discontinuation of test article or withdrawal from the study, if applicable

The participant record is the eCRF or an external record. The author of an entry in the participant record must be identifiable. The first point of entry is considered to be the source record.

Adverse event notes must be reviewed and initialed by the Investigator.

## 16. DATA MANAGEMENT

#### 16.1. Access to Source Data/Document

The Investigator/Institution will permit trial-related monitoring, audits, IEC/IRB review and regulatory inspection(s) by providing direct access to source data/documents. Should the clinical site be contacted for an audit by an IEC/IRB or regulatory authority, JJVC must be contacted and notified in writing within 24 hours.

## 16.2. Confidentiality of Information

Information concerning the investigational product and patent application processes, scientific data or other pertinent information is confidential and remains the property of JJVC. The Investigator may use this information for the purposes of the study only. It is understood by the Investigator that JJVC will use information developed in this clinical study in connection with the development of the investigational product and therefore may disclose it as required to other clinical investigators and to regulatory agencies. In order to allow the use of the information derived from this clinical study, the Investigator understands that he/she has an obligation to provide complete test results and all data developed during this study to the Sponsor.

## 16.3. Data Quality Assurance

Steps will be taken to ensure the accuracy and reliability of data, including the selection of qualified investigators and appropriate clinical sites and review of protocol procedures with the Principal Investigator. The Principal Investigator, in turn, must ensure that all Sub-Investigators and clinical site personnel are familiar with the protocol and all study-specific procedures and have appropriate knowledge of the study article.

Training on case report form completion will be provided to clinical site personnel before the start of the study. The Sponsor will review case report forms for accuracy and completeness remotely during the conduct of the study, during monitoring visits, and after transmission to data management. Any data discrepancies will be resolved with the Investigator or designee, as appropriate.

Quality Assurance representatives from JJVC may visit clinical sites to review data produced during the study and to access compliance with applicable regulations pertaining to the conduct of clinical trials. The clinical sites will provide direct access to study-related source data/documents and reports for the purpose of monitoring and auditing by JJVC and for inspection by local and regulatory authorities.

## 17. MONITORING

The study monitors will maintain close contact with the Principal Investigator and the Investigator's designated clinical site personnel. The monitor's responsibilities will include:

- Ensuring that the investigation is being conducted according to the protocol, any subsequent amendments, and regulatory requirements are maintained
- Ensuring the rights and wellbeing of Subjects are protected
- Ensuring adequate resources, including facilities, laboratories, equipment, and qualified clinical site personnel
- Ensuring that protocol deviations are documented with corrective action plans, as applicable
- Ensuring that the clinical site has sufficient test article and supplies
- Clarifying questions regarding the study
- Resolving study issues or problems that may arise
- Reviewing of study records and source documentation verification in accordance with the monitoring plan

#### 18. ETHICAL AND REGULATORY ASPECTS

## 18.1. Study-Specific Design Considerations

Potential Subjects will be fully informed of the risks and requirements of the study and, during the study, Subjects will be given any new information that may affect their decision to continue participation. Subjects will be told that their consent to participate in the study is voluntary and may be withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Only Subjects who are fully able to understand the

risks, benefits, and potential adverse events of the study, and provide their consent voluntarily will be enrolled.

## 18.2. Investigator Responsibility

The Principal Investigator is responsible for ensuring that the clinical study is performed in accordance with the signed agreement, the investigational plan, Section 4 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements. GCP is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human Subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of study Subjects are protected, consistent with the principles of the Declaration of Helsinki 64<sup>th</sup> WMA General Assembly 2013<sup>3</sup> and that the clinical study data are credible. The Investigator must maintain clinical study files in accordance with Section 8 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements.

# 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB)

Before the start of the study, the Investigator (or Sponsor when applicable) will provide the IEC/IRB with current and complete copies of the following documents (where applicable):

- Final protocol and, if applicable, amendments
- Sponsor-approved informed consent form (and any other written materials to be provided to the Subjects)
- Investigator's Brochure (or equivalent information) and amendments
- Sponsor-approved participant recruitment materials
- Information on compensation for study-related injuries or payment to Subjects for participation in the study
- Investigator's curriculum vitae, clinical licenses, or equivalent information (unless not required, as documented by IEC/IRB)
- Information regarding funding, name of the Sponsor, institutional affiliations, other potential conflicts of interest, and incentives for Subjects
- Any other documents that the IEC/IRB requests to fulfill its obligation

This study will be undertaken only after IEC/IRB has given full approval of the final protocol, amendments (if any), the informed consent form, applicable recruiting materials, and participant compensation programs, and the Sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the documents being approved.

During the study, the Investigator (or Sponsor when applicable) will send the following documents to the IEC/IRB for their review and approval, where appropriate:

- Protocol amendments
- Revision(s) to informed consent form and any other written materials to be provided to Subjects
- If applicable, new or revised participant recruitment materials approved by the Sponsor
- Revisions to compensation for study-related injuries or payment to Subjects for participation in the study
- Investigator's Brochure amendments or new edition(s)

- Summaries of the status of the study (at least annually or at intervals stipulated in guidelines of the IEC/IRB)
- Reports of adverse events that are serious, unanticipated, and associated with the test articles, according to the IRB's requirements
- New information that may adversely affect the safety of the Subjects or the conduct of the study
- Major protocol deviations as required by the IEC/IRB
- Report of deaths of Subjects under the Investigator's care
- Notification if a new Investigator is responsible for the study at the clinical site
- Any other requirements of the IEC/IRB

For protocol amendments that increase participant risk, the amendment and applicable informed consent form revisions must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will review and reapprove this clinical study. This request should be documented in writing.

At the end of the study, the Investigator (or Sponsor where required) will notify the IEC/IRB about the study completion. Documentation of this notification must be retained at the clinical site and a copy provided to the CRO or Sponsor as applicable.

#### 18.4. Informed Consent

Each participant must give written consent according to local requirements after the nature of the study has been fully explained. The consent form must be signed before performance of any study-related activity. The consent form that is used must be approved by both the Sponsor and by the reviewing IEC/IRB. The informed consent is in accordance with principles that originated in the Declaration of Helsinki,<sup>3</sup> current ICH<sup>2</sup> and ISO 14155<sup>1</sup> guidelines, applicable regulatory requirements, and Sponsor Policy.

Before entry into the study, the Investigator or an authorized member of the clinical site personnel must explain to potential participant the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort it may entail. Subjects will be informed that their participation is voluntary and that they may withdraw consent to participate at any time.

The participant will be given sufficient time to read the informed consent form and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the participant's dated signature. After having obtained the consent, a copy of the informed consent form must be given to the participant.

## 18.5. Privacy of Personal Data

The collection, processing and disclosure of personal data and medical information related to the Study Subject, and personal data related to Principal Investigator and any clinical site personnel (e.g., name, clinic address and phone number, curriculum vitae) is participant to compliance with the Health Information Portability and Accountability Act (HIPAA) in the United States<sup>5</sup> and other applicable personal data protection and security laws and regulations. Appropriate measures will be employed to safeguard these data, to maintain the confidentiality of the person's related health and medical information, to properly inform the concerned persons about the collection and processing of their personal data, to grant them reasonable access to their personal data and to prevent access by unauthorized persons.

All information obtained during the course of the investigation will be regarded as confidential. All personal data gathered in this trial will be treated in strictest confidence by Investigators, monitors, Sponsor's personnel and IEC/IRB. No data will be disclosed to any third party without the express permission of the participant concerned, with the exception of Sponsor personnel (monitor, auditor), IEC/IRB and regulatory organizations in the context of their investigation related activities that, as part of the investigation will have access to the CRFs and participant records.

The collection and processing of personal data from Subjects enrolled in this study will be limited to those data that are necessary to investigate the efficacy, safety, quality, and utility of the investigational product(s) used in this study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations.

The Sponsor ensures that the personal data will be:

- processed fairly and lawfully
- collected for specified, explicit, and legitimate purposes and not further processed in a way incompatible with these purposes
- adequate, relevant, and not excessive in relation to said purposes
- accurate and, where necessary, kept current

Explicit consent for the processing of personal data will be obtained from the participating participant before collection of data. Such consent should also address the transfer of the data to other entities and to other countries.

The participant has the right to request through the Investigator access to his personal data and the right to request rectification of any data that are not correct or complete. Reasonable steps should be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration must be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of study Subjects confidential.

#### 19. STUDY RECORD RETENTION

In compliance with the ICH/GCP guidelines,<sup>2</sup> the Investigator/Institution will maintain all CRFs and all participant records that support the data collected from each participant, as well as all study documents as specified in ICH/GCP<sup>2</sup> and all study documents as specified by the applicable regulatory requirement(s). The Investigator/Institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained for a minimum of 25 years, and at least two (2) years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least two (2) years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or instructed by the Sponsor. It is the responsibility of the Sponsor to inform the Investigator/Institution as to when these documents no longer need to be retained.

If the responsible Investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the Investigator relocate or dispose of any study documents before having obtained written approval from the Sponsor.

If it becomes necessary for the Sponsor or the appropriate regulatory authority to review any documentation relating to this study, the Investigator must permit access to such reports. If the Investigator has a question regarding retention of study records, he/she should contact JJVC.

## 20. FINANCIAL CONSIDERATIONS

Remuneration for study services and expenses will be set forth in detail in the Clinical Research Agreement. The Research Agreement will be signed by the Principal Investigator and a JJVC management representative prior to study initiation.

JJVC reserves the right to withhold remuneration for costs associated with protocol violations such as:

- Continuing an ineligible participant in the study
- Scheduling a study visit outside the participant's acceptable visit range

JJVC reserves the right to withhold final remuneration until all study related activities have been completed, such as:

- Query resolution
- Case Report Form signature
- Completion of any follow-up action items

#### 21. PUBLICATION

This study will be registered on ClinicalTrials.gov by the sponsor.

#### 22. REFERENCES

- 1. ISO 14155:2011: Clinical Investigation of Medical Devices for Human Subjects Good Clinical Practice. Available at: https://www.iso.org/standard/45557.html
- 2. International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP). Available at: <a href="http://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html">http://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html</a>
- 3. Declaration of Helsinki Ethical principles for Medical Research Involving Human Subjects. Available at: <a href="https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-Subjects/">https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-Subjects/</a>
- 4. United States (US) Code of Federal Regulations (CFR). Available at: <a href="https://www.gpo.gov/fdsys/browse/collectionCfr.action?collectionCode=CFR">https://www.gpo.gov/fdsys/browse/collectionCfr.action?collectionCode=CFR</a>
- 5. Health Information Portability and Accountability Act (HIPAA). Available at: <a href="https://www.hhs.gov/hipaa/for-professionals/privacy/index.html">https://www.hhs.gov/hipaa/for-professionals/privacy/index.html</a>
- 6. Kenward MG and Roger JH. Small Sample Inference for Fixed Effects from Restricted Maximum Likelihood. *Biometrics*. 1997; 53:983–997.

# APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES) AND QUEST/QUANT QUESTIONNAIRES:







10



24

Protocol 5945
25







Confidential



## APPENDIX B: PATIENT INSTRUCTION GUIDE

Will be provided separately

## APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT)

IMPORTANT: Please read carefully and keep this information for future use.

This Package Insert and Fitting Instruction Guide is intended for the Eye Care Professional, but should be made available to patients upon request.

The Eye Care Professional should provide the patient with the appropriate instructions that pertain to the patient's prescribed lenses. Copies are available for download at www.acuvue.com.



1-DAY ACUVUE® MOIST Brand Contact Lenses 1-DAY ACUVUE® MOIST Brand Contact Lenses for ASTIGMATISM 1-DAY ACUVUE® MOIST Brand MULTIFOCAL Contact Lenses

> etafilcon A Soft (hydrophilic) Contact Lenses Visibility Tinted with UV Blocker for Daily Disposable Wear



Quity CAUTION: U.S. Federal law restricts this device to sale by or on the order of a licensed practitioner.

CR-5945, V9.0




## SYMBOLS KEY

The following symbols may appear on the label or packaging:

| SYMBOL | DEFINITION |
|------------|-----------------------------------------------------|
| (li | Consult Instructions for Use |
| *** | Manufacturer |
| سا | Date of Manufacture |
| $\square$ | Use By Date (expiration date) |
| LOT | Batch Code |
| STERILE | Sterilized Using Steam Heat |
| 2 | Do Not Re-Use (Single Use) |
| <b>₩</b> ♦ | Lens Orientation Correct |
| ₩ X | Lens Orientation Incorrect (Lens Inside Out) |
| C€<br>0086 | Quality System Certification Symbol |
| 0 | Fee Paid for Waste Management |
| EC REP | Authorized Representative in the European Community |

Visit www.acuvue.com/guides for additional information about symbols.

## DESCRIPTION

1-DAY ACUVUE® MOIST Brand Contact Lenses, 1-DAY ACUVUE® MOIST Brand Contact Lenses for ASTIGMATISM, and 1-DAY ACUVUE® MOIST Brand MULTIFOCAL Contact Lenses are soft (hydrophilic) contact lenses available as spherical, toric, or multifocal lenses, and include LACREON® Technology.

The lens material (etaflicon A) is a copolymer of 2-hydroxyethyl methacrylate and methacrylic acid cross-linked with 1, 1, 1-trimethylol propane trimethacrylate and ethylene glycol dimethacrylate.

2

CR-5945, V9.0


The lenses are tinted blue using Reactive Blue Dye #4 to make the lenses more visible for handling. A benzotriazole UV absorbing monomer is used to block UV radiation.

## Lens Properties:

The physical/optical properties of the lens are:

• Specific Gravity (calculated): 0.98 – 1.12 Refractive Index: Light Transmittance: 85% minimum Surface Character: Hydrophilic Water Content: 58% Oxygen Permeability (D/k):

VALUE METHOD

21.4 x 10 11 (cm<sup>2</sup>/sec) Fatt (boundary corrected, edge corrected)

(ml O<sub>2</sub>/ml x mm Hg) @ 35°C

28.0 x 10 <sup>11</sup> (cm<sup>2</sup>/sec) Fatt (boundary corrected, non-edge corrected) (ml O<sub>2</sub>/ml x mm Hg) @ 35°C

## Lens Parameters Ranges:

• Diameter (DIA): 12.0 mm to 15.0 mm Center Thickness: Varies with power Base Curve (BC): 7.85 mm to 10.00 mm Spherical Power (D): -20.00D to +20.00D Cylinder Power (CYL): -0.25D to -10.00D Axis (AXIS): 2.5° to 180° ADD Powers: +0.25D to +4.00D

## **AVAILABLE LENS PARAMETERS**

1-DAY ACUVUE® MOIST Brand Contact Lenses are hemispherical shells of the following dimensions:

Diameter (DIA):

Center Thickness: 0.084 mm to 0.230 mm (varies with power)

CR-5945, V9.0




Base Curve (BC): 8.5 mm, 9.0 mm

-0.50D to -6.00D (in 0.25D increments)

-6.50D to -12.00D (in 0.50D increments) +0.50D to +6.00D (in 0.25D increments)

1-DAY ACUVUE® MOIST Brand Contact Lenses for ASTIGMATISM are hemitoric shells of the following dimensions:

Diameter (DIA): 14.5 mm

Center Thickness: 0.090 mm to 0.189 mm (varies with power)

Base Curve (BC): 8.5 mm

Powers (D): +0.00 to -6.00D (in 0.25D increments)

Cylinders (CYL): -0.75D, -1.25D, -1.75D, -2.25D\* Axis (AXIS): 10° to 180° in 10° increments \*-2.25D cylinder is available in 10°, 20°, 70°, 80°, 90°, 100°, 110°, 160°, 170°, 180° axes only

-6.50D to -9.00D (in 0.50D increments)

Cylinders (CYL): -0.75D, -1.25D, -1.75D, -2.25D\* Axis (AXIS): 10°, 20°, 60°, 70°, 80°, 90°, 100°, 110°,

120°, 160°, 170°, 180°

\*-2.25D cylinder is available in 20°, 90°, 160°, 180°

axes only

+0.25D to +4.00D (in 0.25D increments) Cylinders (CYL): -0.75D, -1.25D, -1.75D

Axis (AXIS): 10°, 20°, 70°, 80°, 90°, 100°, 110°, 160°,

170°, 180°

1-DAY ACUVUE® MOIST Brand MULTIFOCAL Contact Lenses are hemispherical shells of the following dimensions:

Diameter (DIA): 14.3 mm

Center Thickness: 0.084 mm to 0.207 mm (varies with power)

Base Curve (BC): 8.4 mm

Powers (D): +6.00D to -9.00D (in 0.25D increments) Near ADD Powers Low Near ADD (LOW): +1.25D (MAX ADD): Medium Near ADD (MID): +1.75D

High Near ADD (HGH): +2.50D

CR-5945, V9.0




## TRANSMITTANCE CURVES

1-DAY ACUVUE® MOIST Brand Contact Lenses (etaflicon A) Visibility Tinted with UV Blocker vs. 24 yr. old human cornea and 25 yr. old human crystalline lens.



 $^*$ The data are representative measurements taken through the central 3-5 mm portion for the thinnest marketed lens (-3.00D lens, 0.084 mm center thickness).

<sup>1</sup> Lerman, S., Radiant Energy and the Eye, MacMillan, New York, 1980, p. 58, figure 2-21
<sup>2</sup> Waxler, M., Hitchins, V.M., Optical Radiation and Visual Heath, CRC Press, Boca Raton, Florida, 1986, p. 19, figure 5

WARNING: UV absorbing contact lenses are NOT substitutes for protective UV absorbing eyewear, such as UV absorbing goggles or sunglasses because they do not completely cover the eye and surrounding area. The patient should continue to use UV absorbing eyewear as directed.

## **ACTIONS**

In its hydrated state, the contact lens, when placed on the cornea, acts as a refracting medium to focus light rays on the retina.

The UV Blocking for these lenses averages 97% in the UVB range of 280 nm to 315 nm and 82% in the UVA range of 316 nm to 380 nm for the entire power range.

5



NOTE: Long-term exposure to UV radiation is one of the risk factors associated with cataracts. Exposure is based on a number of factors such as environmental conditions (altitude, geography, cloud cover) and personal factors (extent and nature of outdoor activities). UV-Blocking contact lenses help provide protection against harmful UV radiation. However, clinical studies have not been done to demonstrate that wearing UV-Blocking contact lenses reduces the risk of developing cataracts or other eye disorders. The Eye Care Professional should be consulted for more information.

## **INDICATIONS (USES)**

1-DAY ACUVUE® MOIST Brand Contact Lenses are indicated for daily disposable wear for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes who may have 1.00D or less of astigmatism.

1-DAY ACUVUE® MOIST Brand Contact Lenses for ASTIGMATISM are indicated for daily disposable wear for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes who may have 0.50D to 3.00D of astigmatism.

1-DAY ACUVUE® MOIST Brand MULTIFOCAL Contact Lenses are indicated for daily disposable wear for the optical correction of distance and near vision in presbyopic phakic or aphakic persons with non-diseased eyes who may have 4,00D of ADD power or less and 0,75D or less of astigmatism.

The lenses contain a UV Blocker to help protect against transmission of harmful UV radiation to the comea and into the eye.

When prescribed for daily disposable use, no cleaning or disinfection is required. Lenses should be discarded upon removal.

## CONTRAINDICATIONS (REASONS NOT TO USE)

DO NOT USE these lenses when any of the following conditions exist:

- Acute or subacute inflammation or infection of the anterior chamber of the eye.
- Any eye disease, injury, or abnormality that affects the cornea, conjunctiva, or eyelids.
- · Severe insufficiency of lacrimal secretion (dry eye).
- · Corneal hypoesthesia (reduced corneal sensitivity).

6



- Any systemic disease that may affect the eye or be exaggerated by wearing contact lenses.
- Allergic reactions of ocular surfaces or adnexa that may be induced or exaggerated by wearing contact lenses or use of contact lens solutions.
- Ocular irritation due to allergic reactions which may be caused by use
  of contact lens solutions (i.e., rewetting drops) that contain chemicals or
  preservatives (such as mercury, Thimerosal, etc.) to which some people
  may develop an allergic response.
- Any active corneal infection (bacterial, fungal, protozoal, or viral).
- If eyes become red or irritated.

## **WARNINGS**

Patients should be advised of the following warnings pertaining to contact lens wear:

EYE PROBLEMS, INCLUDING CORNEAL ULCERS, CAN DEVELOP RAPIDLY AND LEAD TO LOSS OF VISION. IF THE PATIENT EXPERIENCES:

- Eye Discomfort,
- Excessive Tearing,
- · Vision Changes,
- . Loss of Vision,
- Eye Redness, or
- Other Eye Problems,

THE PATIENT SHOULD BE INSTRUCTED TO IMMEDIATELY REMOVE THE LENSES AND PROMPTLY CONTACT THE EYE CARE PROFESSIONAL.

- When prescribed for daily wear, patients should be instructed not to wear their lenses while sleeping. Clinical studies have shown that when lenses are worn overnight, the risk of ulcerative keratitis is greater than among those who do not wear them overnight.<sup>3</sup>
- Studies have shown that contact lens wearers who are smokers have a higher incidence of adverse reactions than nonsmokers.
- Problems with contact lenses or lens care products could result in serious injury to the eye. Patients should be cautioned that proper use and care of contact lenses and lens care products are essential for the safe use of these products.

7



 The overall risk of ulcerative keratitis may be reduced by carefully following directions for lens care.

<sup>3</sup> New England Journal of Medicine, September 21, 1989; 321 (12), pp. 773-783

#### Specific Instructions for Use and Warnings:

Water Activity

Instruction for Use

Do not expose contact lenses to water while wearing them.

#### WARNING:

Water can harbor microorganisms that can lead to severe infection, vision loss, or blindness. If lenses have been submersed in water when participating in water sports or swimming in pools, hot tubs, lakes, or oceans, the patient should be instructed to discard them and replace them with a new pair. The Eye Care Professional should be consulted for recommendations regarding wearing lenses during any activity involving water.

#### **PRECAUTIONS**

### Special Precautions for Eye Care Professionals:

 Due to the small number of patients enrolled in clinical investigation of lenses, all refractive powers, design configurations, or lens parameters available in the lens material are not evaluated in significant numbers. Consequently, when selecting an appropriate lens design and parameters, the Eye Care Professional should consider all characteristics of the lens that can affect lens performance and ocular health, including oxygen permeability, wettability, central and peripheral thickness, and optic zone diameter.

The potential impact of these factors on the patient's ocular health should be carefully weighed against the patient's need for refractive correction; therefore, the continuing ocular health of the patient and lens performance on the eye should be carefully monitored by the prescribing Eye Care Professional.

 Patients who wear these lenses to correct presbyopia using monovision (or modified monovision using 1-DAY ACUVUE® MOIST Brand MULTIFOCAL) may not achieve the best corrected visual acuity for either far or near vision. Visual requirements vary with the individual and should be considered when selecting the most appropriate type of lens for each patient.

Q



- Fluorescein, a yellow dye, should not be used while the lenses are on the eyes. The lenses absorb this dye and become discolored. Whenever fluorescein is used in eyes, the eyes should be flushed with a sterile saline solution that is recommended for in-eye use.
- Eye Care Professionals should instruct the patient to remove lenses immediately if the eyes become red or irritated.

# Eye Care Professionals should carefully instruct patients about the following care regimen and safety precautions.

#### **Handling Precautions:**

- Before leaving the Eye Care Professional's office, the patient should be able to promptly remove the lenses or should have someone else available who can remove the lenses for him or her.
- DO NOT use if the sterile blister package is opened or damaged.
- Always wash and rinse hands before handling lenses. Do not get cosmetics, lotions, soaps, creams, deodorants, or sprays in the eyes or on the lenses. It is best to put on lenses before putting on makeup.
- DO NOT touch contact lenses with the fingers or hands if the hands are
  not free of foreign materials, as microscopic scratches of the lenses may
  occur, causing distorted vision and/or injury to the eye.
- Carefully follow the handling, insertion, removal, and wearing instructions in the Patient instruction Guide for these lenses and those prescribed by the Eye Care Professional.
- · Always handle lenses carefully and avoid dropping them.
- Never use tweezers or other tools to remove lenses from the lens container. Slide the lens up the side of the bowl until it is free of the container.
- Do not touch the lens with fingernails.

## Lens Wearing Precautions:

- If the lens sticks (stops moving) on the eye, follow the recommended directions in "Care for Sticking (Non-Moving) Lenses." The lens should move freely on the eye for the continued health of the eye. If nonmovement of the lens continues, the patient should be instructed to immediately consult his or her Eye Care Professional.
- Never wear lenses beyond the period recommended by the Eye Care Professional.

a



- The patient should be advised to never allow anyone else to wear their lenses. They have been prescribed to fit their eyes and to correct their vision to the degree necessary. Sharing lenses greatly increases the chance of eye infections.
- If aerosol products, such as hairspray, are used while wearing lenses, exercise caution and keep eyes closed until the spray has settled.
- · Avoid all harmful or irritating vapors and fumes while wearing lenses.

#### Lens Care Precautions:

 The patient should be informed that no cleaning or disinfection is needed when lenses are worn for daily disposable wear. Patients should always dispose of lenses when removed and have spare lenses or spectacles available.

## Other Topics to Discuss with Patients:

- Always contact the Eye Care Professional before using any medicine in the eyes.
- Certain medications, such as antihistamines, decongestants, diuretics, muscle relaxants, tranquilizers, and those for motion sickness may cause dryness of the eye, increased lens awareness, or blurred vision. Should such conditions exist, proper remedial measures should be prescribed.
- Oral contraceptive users could develop visual changes or changes in lens tolerance when using contact lenses. Patients should be cautioned accordingly.
- As with any contact lens, follow-up visits are necessary to assure the continuing health of the patient's eyes. The patient should be instructed as to a recommended follow-up schedule.

## Who Should Know That the Patient is Wearing Contact Lenses?

- Patients should inform all doctors (Health Care Professionals) about being a contact lens wearer.
- Patients should always inform their employer of being a contact lens wearer. Some jobs may require use of eye protection equipment or may require that the patient not wear contact lenses.

10



## **ADVERSE REACTIONS**

The patient should be informed that the following problems may occur when wearing contact lenses:

- The eye may burn, sting, and/or itch.
- There may be less comfort than when the lens was first placed on the eye.
- There may be a feeling of something in the eye (foreign body, scratched area).
- There may be the potential for some temporary impairment due to peripheral infiltrates, peripheral corneal ucers, or corneal erosion. There may be the potential for other physiological observations, such as local or generalized edema, corneal neovascularization, corneal staining, injection, tarsal abnormalities, iritis, and conjunctivitis, some of which are clinically acceptable in low amounts.
- There may be excessive watering, unusual eye secretions, or redness of the eve.
- Poor visual acuity, blurred vision, rainbows or halos around objects, photophobia, or dry eyes may also occur if the lenses are worn continuously or for too long a time.

The patient should be instructed to conduct a simple 3-part self-examination at least once a day. They should ask themselves:

- How do the lenses feel on my eyes?
- How do my eyes look?
- Have I noticed a change in my vision?

If the patient reports any problems, he or she should be instructed to IMMEDIATELY REMOVE THE LENS. If the problem or discomfort stops, the patient should discard the lens and place a new fresh lens on the eye.

If after inserting the new lens, the problem continues, the patient should be directed to IMMEDIATELY REMOVE THE LENS AND CONTACT HIS OR HER EYE CARE PROFESSIONAL.

The patient should be advised that when any of the above symptoms occur, a serious condition such as infection, corneal ulcer, neovascularization, or iritis may be present. He or she should be instructed to seek immediate professional identification of the problem and prompt treatment to avoid serious eye damage.

11



## **GENERAL FITTING GUIDELINES**

#### A. Patient Selection

Patients selected to wear these lenses should be chosen based on:

- · Motivation to wear lenses
- Ability to follow instructions regarding lens wear
- General health
- Ability to adequately handle and care for the lenses
- · Ability to understand the risks and benefits of lens wear

Patients who do not meet the above criteria should not be provided with contact language.

#### B. Pre-fitting Examination

Initial evaluation of the patient should begin with a thorough case history to determine if there are any contraindications to contact lens wear. During the case history, the patient's visual needs and expectations should be determined as well as an assessment of their overall ocular, physical, and mental health.

Preceding the initial selection of trial contact lenses, a comprehensive ocular evaluation should be performed that includes, but is not limited to, the measurement of distance and near visual acuity, distance and near refractive prescription (including determining the preferred reading distance for presbyopes), keratometry, and biomicroscopic evaluation.

Based on this evaluation, if it is determined that the patient is eligible to wear these lenses, the Eye Care Professional should proceed to the lens fitting instructions as outlined below.

## C. Initial Power Determination

A spectacle refraction should be performed to establish the patient's baseline refractive status and to guide in the selection of the appropriate lens power. Remember to compensate for vertex distance if the refraction is greater than ±4,00D.

## D. Base Curve Selection (Trial Lens Fitting)

The following trial lenses should be selected for patients regardless of keratometry readings. However, comeal curvature measurements should be performed to establish the patient's baseline ocular status.

12



- 1-DAY ACUVUE® MOIST: 8.5 mm/14.2 mm
- 1-DAY ACUVUE® MOIST for ASTIGMATISM: 8.5 mm/14.5 mm
- 1-DAY ACUVUE® MOIST MULTIFOCAL: 8.4 mm/14.3 mm

The trial lens should be placed on each of the patient's eyes and evaluated after the patient has adjusted to the lenses.

## 1. Criteria of a Property Fit Lens

A properly fit lens will center and completely cover the cornea (i.e., no limbal exposure), have sufficient movement to provide tear exchange under the contact lens with the blink, and be comfortable. The lens should move freely when manipulated digitally with the lower lid, and then return to its properly centered position when released.

## 2. Criteria of a Flat Fitting Lens

A flat fitting lens may exhibit one or more of the following characteristics: decentration, incomplete comeal coverage (i.e., limbal exposure), excessive movement with the blink and/or edge standoff. If the lens is judged to be flat fitting, it should not be dispensed to the patient.

#### 3. Criteria of a Steep Fitting Lens

A steep fitting lens may exhibit one or more of the following characteristics: insufficient movement with the blink, conjunctival indentation, and resistance when pushing the lens up digitally with the lower lid. If the lens is judged to be steep fitting, it should not be dispensed to the patient.

If the initial trial base curve is judged to be flat or steep fitting, the alternate base curve, if available, should be trial fit and evaluated after the patient has adjusted to the lens. The lens should move freely when manipulated digitally with the lower lid, and then return to a properly centered position when released. If resistance is encountered when pushing the lens up, the lens is fitting tightly and should not be dispensed to the patient.

## E. Final Lens Power (Spherical)

A spherical over-refraction should be performed to determine the final lens power after the lens fit is judged acceptable. The spherical over-refraction should be combined with the trial lens power to determine the final lens prescription. The patient should experience good visual acuity with the correct lens power unless there is excessive residual astigmatism.

13



| Example 1 | |
|----------------------------|--------|
| Diagnostic lens: | -2.00D |
| Spherical over-refraction: | -0.25D |
| Final lens power: | -2.25D |
| Example 2 | |
| Diagnostic lens: | -2.00D |
| Spherical over-refraction: | +0.25D |

If vision is acceptable, perform a slit lamp examination to assess adequate fit (centration and movement). If the fit is acceptable, dispense the lenses and instruct the patient to return in one week for reassessment (see **PATIENT MANAGEMENT** section).

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

## **TORIC FITTING GUIDELINES**

Although most aspects of the fitting procedure are identical for all types of soft contact lenses, including toric lenses, there are some additional steps and/or rules to follow to assure the proper fit of toric lenses.

The only new steps you must follow in prescribing 1-DAY ACUVUE® MOIST for ASTIGMATISM are that you must determine the stability, repeatability, and drift angle of the lens axis so that you can prescribe the correct lens axis for the nation!

## A. How to Determine Lens Cylinder and Axis Orientation

## 1. Locate the Orientation Marks

To help determine the proper orientation of the toric lens, you'll find two primary marks approximately 1 mm from the lens edge representing the vertical position on opposite ends of the lens at 6 and 12 o'clock (Fig. 1). Because of the lens' ballasting system, either mark can represent the vertical position – there is no "top" and "bottom" as in a prism-ballasted lens. You don't need to view both marks to assess orientation; simply look for the 6 o'clock mark as you would with a prism-ballasted lens.

14





You'll need a slit lamp biomicroscope with a 1 to 2 mm parallelepiped beam to highlight the marks when the lens is fitted to the eye. There are a number of techniques you can use to improve the visibility of the 6 o'clock mark. Using a parallelepiped beam and medium magnification (10x or 15x), slowly pan down the lens, looking just below the direct illumination at the retroilluminated area. Backlighting the mark this way should make it more visible. Sometimes manipulating the lower lid may be necessary to uncover the mark.

#### 2. Observe Lens Rotation and Stability

Observe the position and stability of the "bottom" mark. It usually stabilizes at the 6 o'clock position. If it does, calculation of the lens power will be straightforward. The 6 o'clock position is not a "must"; however, the absolute requirement is that the axis position be stable and repeatable.

The mark may stabilize somewhat left or right (drift) of the vertical meridian and still enable you to fit a toric lens for that eye, as long as the lens always returns to the same "drift axis" position after settling. The deviation can be compensated for in the final prescription. Your objective is to ensure that whatever position the initial lens assumes near 6 o'clock, this position must be stable and repeatable. With full eye movement or heavy blink, you may see the marks swing away, but they must return quickly to the original stable position. If the lens does not return quickly, you may need to select a different lens.

## 3. Assessing Rotation

Imagine the eye as a clock dial and every hour represents a 30° interval. If the orientation mark of the initial lens stabilizes somewhat left or right of the vertical position, the final lens will orient on the eye with the same deviation. You can use an axis reticule in the slit lamp or use a line-scribed lens in a spectacle trial frame to measure or estimate the "drift angle" of the cylinder axis

To compensate for this "drift," measure or estimate the "drift," then add or subtract it from the refractive axis to determine the correct cylinder axis. Use the LARS (Left Add, Right Subtract) method to determine which direction to compensate.

15


#### B. Final Lens Power

When the diagnostic lens has its axis aligned in the same meridian as the patient's refractive axis, a spherocylindrical over-refraction may be performed and visual acuity determined. However, in the case of crossed axes, such as when the diagnostic lens axis is different from the spectacle cylinder axis, it is not advisable to perform a full spherocylindrical over-refraction because of the difficulty in computing the resultant power. A spherical over-refraction without cylinder refraction may be performed.

If the required cylinder correction falls between two available cylinder powers, it is recommended to prescribe the lower cylinder power lens. See below for instructions on how to determine the final lens power.

#### 1. For the Sphere

If sphere alone or combined sphere and cylinder Rx > 4.00D, compensate for vertex distance. If sphere alone or combined sphere and cylinder Rx  $\leq$   $\pm$ 4.00D, vertex compensation is not necessary.

#### 2. For the Cylinder

Adjust the axis by the drift angle using the LARS method. Choose a cylinder that is  $\leq 0.50D$  from the refractive cylinder.

## 3. Case Examples

## Example 1

Manifest (spectacle) refraction:

O.D. -2.50D / -1.25D x 180° 20/20 O.S. -2.00D / -1.00D x 180° 20/20

Choose a diagnostic lens for each eye with axis  $180^\circ$ . Place the lens on each eye and allow a minimum of 3 minutes for it to equilibrate, based on the patient's initial response to the lens. If the lens has not yet stabilized, recheck until stable.

Check the orientation of the axis mark. If the bottom axis mark is in the 6 o'clock position on both eyes, choose the appropriate cylinder as listed previously. If the lens has not yet stabilized, recheck until stable.

Here is the Rx prescribed:

O.D. -2.50D / -1.25D x 180°

O.S. -2.00D / -0.75D x 180°

16



## Example 2

Manifest (spectacle) refraction: O.D. -3.00D / -1.00D x 90° 20/20 O.S. -4.75D / -2.00D x 90° 20/20

Choose diagnostic lenses of -3.00D / -0.75D x 90° for the right eye and -4.50D / -1.75D x 90° for the left eye, the nearest lenses available to the spherical power and axis needed. For the left eye, since the manifest refraction called for -4.75D, compensating for vertex distance the sphere is reduced by 0.25D to -4.50D. The cylinder power will be -1.75D. Place the lens on each eye and allow a minimum of 3 minutes for it to equilibrate, based on the patient's initial response to the lens. If the lens has not yet stabilized, recheck until stable.

#### Right Eye

The orientation mark on the right lens rotates left from the 6 o'clock position by  $10^{\circ}$  and remains stable in this position. Compensation for this rotation should be done as follows:

Compensate the 10° axis drift by adding it to the manifest refraction axis.

Here is the Rx prescribed: O.D. -3.00D / -0.75D x 100°

## Left Eye

The orientation mark on the left lens rotates right from the 6 o'clock position by 10° and remains stable in this position. Compensation for this rotation should be done as follows:

Compensate for the 10° axis drift by subtracting it from the manifest refraction axis.

Here is the Rx prescribed:

O.S. -4.50D / -1.75D x 80°

If vision is acceptable, perform a slit lamp examination to assess adequate fit (centration and movement). If fit is acceptable, dispense the lenses instructing the patient to return in one week for reassessment (see PATIENT MANAGEMENT section).

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.


#### **MULTIFOCAL FITTING GUIDELINES**

#### A. Presbyopic Needs Assessment & Patient Education

Multifocal contact lenses may produce compromise to vision under certain circumstances and the patient should understand that they might not find their vision acceptable in specific situations (i.e., reading a menu in a dim restaurant, driving at night in rainy/foggy conditions, etc.). Therefore, caution should be exercised when the patient is wearing the correction for the first time until they are familiar with the vision provided in visually challenging environments. Occupational and environmental visual demands should be considered. If the patient requires critical visual acuity and stereopsis, it should be determined by trial whether this patient can function adequately with 1-DAY ACUVUE® MOIST MULTIFOCAL. Wearing these lenses may not be optimal for activities such as:

- Visually demanding situations such as operating potentially dangerous machinery or performing other potentially hazardous activities; and
- Driving automobiles (e.g., driving at night). Patients who cannot meet
  their state driver's license requirements with the 1-DAY ACUVUE® MOIST
  MULTIFOCAL should be advised to not drive with this correction, OR may
  require that additional over-correction be prescribed.

1-DAY ACUVUE® MOIST MULTIFOCAL is not recommended for patients who have -1.00D or greater of refractive cylinder as this level of uncorrected cylinder may lead to additional visual compromise. These lenses are available in the following ADD powers:

- Lens "LOW" = low near ADD lens (Max ADD +1.25)
- Lens "MID" = medium near ADD lens (Max ADD +1.75)
- Lens "HGH" = high near ADD lens (Max ADD +2.50)

#### **B. Initial Power Determination**

A spectacle refraction should be performed to establish the patient's baseline refractive status and to guide in the selection of the appropriate lens power. Remember to compensate for vertex distance if the refraction is greater than  $\pm 4.00D$ . Determine the spherical equivalent distance prescription for a multifocal patient. Determine the eye dominance using one of the methods below:

18



Method 1 Determine which eye is the "sighting eye." Have the patient point to an object at the far end of the room. Cover one eye. If the patient is still pointing directly at the object, the eye being used is the dominant (sighting) eye.

Method 2 Determine which eye does not accept added plus power. Place a +1.00D hand-held trial lens in front of one eye and then the other while the distance refractive error correction is in place for both eyes while the patient is viewing the distance visual acuity chart. The eye with the plus over it that the patient notices the greatest reduction in vision is determined to be the dominant eye.

#### C. Select the Initial Trial Lens

- 1. For each eye, select the trial lens distance power that is closest to the patient's distance spherical equivalent. Remember to compensate for vertex distance if the refraction is greater than  $\pm 4.00D$ .
- 2. Select the near power of the lens based on the patients ADD range as
  - ADD: +0.75D to +1.25D use a low near ADD (LOW) lens on each eye
  - ADD: +1.50D to +1.75D use a medium near ADD (MID) lens on each
  - ADD: +2.00D to +2.50D use a medium near ADD (MID) on the dominant eye and a high near ADD (HGH) lens on the non-dominant
- 3. Allow the lenses to settle for a minimum of 10 minutes.
- 4. Assess distance and near vision binocularly and monocularly.
- 5. Demonstrate the vision under various lighting conditions (normal and decreased illumination) and at distance, intermediate, and near.
- 6. Make adjustments in power as necessary based on the distance overrefraction. The use of hand-held trial lenses is recommended. Check the impact on distance and near vision.
- 7. If vision is still unacceptable, make adjustments in power as necessary (see "Multifocal Troubleshooting" below). If distance and near vision are acceptable, perform a slit lamp examination to assess adequate fit (centration and movement). If fit is acceptable, dispense the lenses instructing the patient to return in one week for reassessment (see PATIENT MANAGEMENT section).



#### D. Multifocal Troubleshooting

#### Unacceptable Near Vision

If it has been determined that no change is required based on the overrefraction, then add +0.25D to the spherical power of the non-dominant eye.

#### **Unacceptable Distance Vision**

If it has been determined that no change is required based on the overrefraction, then make the changes as listed below:

- If the patient is wearing two "LOW" ADD lenses, change the dominant eye to a 1-DAY ACUVUE® MOIST sphere lens with a power equal to the spherical equivalent distance prescription.
- If the patient is wearing two "MID" ADD lenses, change the ADD power in the dominant eye to the "LOW" ADD power.
- If the patient is wearing a "MID" ADD lens in the dominant eye and a "HGH" ADD lens in the non-dominant eye, change the non-dominant eye to a "MID" ADD lens and add +0.25D to the distance power.

#### E. Adaptation

Visually demanding situations should be avoided during the initial wearing period. A patient may at first experience some mild blurred vision, dizziness, headaches and a feeling of slight imbalance. You should explain the adaptational symptoms to the patient. These symptoms may last for a brief minute or for several weeks. The longer these symptoms persist, the poorer the prognosis for successful adaptation.

To help in the adaptation process, the patient can be advised to first use the lenses in a comfortable, familiar environment such as in the home.

Some patients feel that automobile driving performance may not be optimal during the adaptation process. This is particularly true when driving at night. Before driving a motor vehicle, it may be recommended that the patient be a passenger first to make sure that their vision is satisfactory for operating an automobile. During the first several weeks of wear (when adaptation is occurring), it may be advisable for the patient to only drive during optimal driving conditions. After adaptation and success with these activities, the patient should be able to drive under other conditions with caution.

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

20



#### MONOVISION FITTING GUIDELINES

#### A. Patient Selection

#### 1. Monovision Needs Assessment

For a good prognosis, the patient should have adequately corrected distance and near visual acuity in each eye. The amblyopic patient or the patient with significant astigmatism (greater than 1.00D) in one eye may not be a good candidate for monovision correction with these lenses.

Occupational and environmental visual demands should be considered. If the patient requires critical vision (visual acuity and stereopsis), it should be determined by trial whether this patient can function adequately with monovision correction. Monovision contact lens wear may not be optimal for activities such as:

- Visually demanding situations such as operating potentially dangerous machinery or performing other potentially hazardous activities; and
- Driving automobiles (e.g., driving at night). Patients who cannot meet
  their state driver's license requirements with monovision correction
  should be advised to not drive with this correction, OR may require that
  additional over-correction be prescribed.

#### 2. Patient Education

All patients do not function equally well with monovision correction. Patients may not perform as well for certain tasks with this correction as they have with spectacles (multifocal, bifocal, trifocal, readers, progressives). Each patient should understand that monovision, as well as other presbyopic alternatives, can create a vision compromise that may reduce visual acuity and depth perception for distance and near tasks. Therefore, caution should be exercised when the patient is wearing the correction for the first time until they are familiar with the vision provided in visually challenging environments (e.g., reading a menu in a dimly lit restaurant, driving at night in rainy/foggy conditions, etc.). During the fitting process, it is necessary for the patient to realize the disadvantages as well as the advantages of clear near vision, and straight ahead and upward gaze that monovision contact lenses provide.

21



#### B. Eye Selection

#### 1. Ocular Preference Determination Methods

Generally, the non-dominant eye is corrected for near vision. The following two methods for eye dominance can be used.

Method 1 Determine which eye is the "sighting eye." Have the patient point to an object at the far end of the room. Cover one eye. If the patient is still pointing directly at the object, the eye being used is the dominant (sighting) eye.

Method 2 Determine which eye will accept the added power with the least reduction in vision. Place a hand-held trial lens equal to the spectacle near ADD in front of one eye and then the other while the distance refractive error correction is in place for both eyes. Determine whether the patient functions best with the near ADD lens over the right or left eye.

#### 2. Other Eye Selection Methods

Other methods include the "Refractive Error Method" and the "Visual Demands Method."

#### Refractive Error Method

For anisometropic correction, it is generally best to fit the more hyperopic (less myopic) eye for distance and the more myopic (less hyperopic) eye for near.

#### Visual Demands Method

Consider the patient's occupation during the eye selection process to determine the critical vision requirements. If a patient's gaze for near tasks is usually in one direction, correct the eye on that side for near.

Example: A secretary who places copy to the left side of the desk will function best with the near lens on the left eye.

#### C. Special Fitting Characteristics

#### 1. Unilateral Vision Correction

There are circumstances where only one contact lens is required. As an example, an emmetropic patient would only require a near lens, whereas a bilateral myope would require corrective lenses on both eyes.

22



#### Examples:

A presbyopic emmetropic patient who requires a +1.75D ADD would have a +1.75D lens on the near eye and the other eye left without correction.

A presbyopic patient requiring a +1.50D ADD who is -2.50D myopic in the right eye and -1.50D myopic in the left eye may have the right eye corrected for distance and the left eye uncorrected for near.

#### 2. Near ADD Determination

Always prescribe the lens power for the near eye that provides optimal near acuity at the midpoint of the patient's habitual reading distance. However, when more than one power provides optimal reading performance, prescribe the least plus (most minus) of the powers.

#### 3. Trial Lens Fitting

A trial fitting is performed in the office to allow the patient to experience monovision correction. Lenses are fit according to the **GENERAL FITTING GUIDELINES** for base curve selection described in this Package Insert.

Case history and a standard clinical evaluation procedure should be used to determine the prognosis. Determine the distance correction and the near correction. Next, determine the near ADD. With trial lenses of the proper power in place, observe the reaction to this mode of correction.

Allow the lenses to settle for about 20 minutes with the correct power lenses in place. Walk across the room and have the patient look at you. Assess the patient's reaction to distance vision under these circumstances. Then have the patient look at familiar near objects such as a watch face or fingernails. Again assess the reaction. As the patient continues to look around the room at both near and distance objects, observe the reactions. Only after these vision tests are completed, should the patient be asked to read print. Evaluate the patient's reaction to large print (e.g., typewritten copy) at first and then graduate to newsprint and finally smaller type sizes.

After the patient's performance under the above conditions is completed, tests of visual acuity and reading ability under conditions of moderately dim illumination should be attempted.

23



An initial unfavorable response in the office, while indicative of a guarded prognosis, should not immediately rule out a more extensive trial under the usual conditions in which a patient functions.

#### 4. Adaptation

Visually demanding situations should be avoided during the initial wearing period. A patient may at first experience some mild blurred vision, dizziness, headaches, and a feeling of slight imbalance. You should explain the adaptational symptoms to the patient. These symptoms may last for a brief minute or for several weeks. The longer these symptoms persist, the poorer the prognosis for successful adaptation.

To help in the adaptation process, the patient can be advised to first use the lenses in a comfortable, familiar environment such as in the home.

Some patients feel that automobile driving performance may not be optimal during the adaptation process. This is particularly true when driving at night. Before driving a motor vehicle, it may be recommended that the patient be a passenger first to make sure that their vision is satisfactory for operating an automobile. During the first several weeks of wear (when adaptation is occurring), it may be advisable for the patient to only drive during optimal driving conditions. After adaptation and success with these activities, the patient should be able to drive under other conditions with caution.

#### D. Other Suggestions

The success of the monovision technique may be further improved by having your patient follow the suggestions below:

- Have a third contact lens (distance power) to use when critical distance viewing is needed.
- Have a third contact lens (near power) to use when critical near viewing is needed.
- Have supplemental spectacles to wear over the monovision contact lenses for specific visual tasks may improve the success of monovision correction. This is particularly applicable for those patients who cannot meet state driver's licensing requirements with monovision correction.
- · Make use of proper illumination when carrying out visual tasks.

24



Monovision fitting success can be improved by the following suggestions:

- Reverse the distance and near eyes if a patient is having trouble adapting.
- Refine the lens powers if there is trouble with adaptation. Accurate lens power is critical for presbyopic patients.
- Emphasize the benefits of clear near vision, and straight ahead and upward gaze with monovision.

The decision to fit a patient with monovision correction is most appropriately left to the Eye Care Professional in conjunction with the patient after carefully considering the patient's needs.

All patients should be supplied with a copy of the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

#### PATIENT MANAGEMENT

- Follow the accepted standard of care in fitting and following up with your patient, e.g., American Optometric Association standard of care.
- Schedule the appropriate follow-up examination.
- Preferably, at the follow-up visits, lenses should have been worn for at least six hours.
- Provide the patient with a copy of the PATIENT INSTRUCTION GUIDE for these lenses, which can be found at www.acuvue.com. REVIEW THESE INSTRUCTIONS WITH THE PATIENT SO THAT HE OR SHE CLEARLY UNDERSTANDS THE PRESCRIBED WEARING AND REPLACEMENT SCHEDULES.

#### WEARING SCHEDULE

The wearing schedule should be determined by the Eye Care Professional. Regular checkups, as determined by the Eye Care Professional, are also extremely important.

Patients tend to over wear the lenses initially. The Eye Care Professional should emphasize the importance of adhering to the initial maximum wearing schedule. Maximum wearing time should be determined by the Eye Care Professional based upon the patient's physiological eye condition, because individual response to contact lenses varies.

25



The maximum suggested wearing time for these lenses is:

| DAY | HOURS |
|-------------|------------------|
| 1 | 6-8 |
| 2 | 8-10 |
| 3 | 10-12 |
| 4 | 12-14 |
| 5 and after | all waking hours |

### REPLACEMENT SCHEDULE

These lenses are indicated for daily disposable wear and should be discarded upon removal.

When disposed of after a single daily use, these lenses may reduce the risk of developing giant papillary conjunctivitis.<sup>4</sup>

When worn as a daily disposable lens, these lenses may provide improved comfort for many patients who experience mild discomfort and itching associated with allergies during contact lens wear, compared to lenses replaced at intervals of greater than 2 weeks.

Clinical research has shown that when worn on a daily disposable basis, these lenses may provide improved comfort for 2 out of 3 patients who reported suffering from discomfort associated with allergies during contact lens wear.

## LENS CARE DIRECTIONS

The Eye Care Professional should review with patients that no cleaning or disinfection is needed with daily disposable lenses. Patients should always dispose of lenses when they are removed and have replacement lenses or spectacles available.

For complete information concerning contact lens handling and care, refer to the PATIENT INSTRUCTION GUIDE for these lenses. Copies are available for download at www.acuvue.com.

#### Care for Sticking (Non-Moving) Lenses

During removal, if the lens sticks to the eye, the patient should be instructed to apply a few drops of the recommended lubricating or rewetting solution

26



<sup>&</sup>lt;sup>4</sup>The CLAO Journal, July 1999, Volume 25, Number 3

directly to the eye and wait until the lens begins to move freely on the eye before removing it. If non-movement of the lens continues after a few minutes, the patient should **immediately** consult the Eye Care Professional.

#### **EMERGENCIES**

The patient should be informed that if chemicals of any kind (household products, gardening solutions, laboratory chemicals, etc.) are splashed into the eyes, the patient should: FLUSH EYES IMMEDIATELY WITH TAP WATER AND IMMEDIATELY CONTACT THE EYE CARE PROFESSIONAL OR VISIT A HOSPITAL EMERGENCY ROOM WITHOUT DELAY.

#### **HOW SUPPLIED**

Each UV-absorbing sterile lens is supplied in a foil-sealed plastic package containing buffered saline solution with povidone. The plastic package is marked with the following:

- 1-DAY ACUVUE® MOIST: base curve, power, diameter, lot number, and expiration date
- 1-DAY ACUVUE® MOIST for ASTIGMATISM: base curve, power, diameter, cylinder, axis, lot number, and expiration date
- 1-DAY ACUVUE® MOIST MULTIFOCAL: base curve, power, diameter, ADD power, lot number, and expiration date

### REPORTING OF ADVERSE REACTIONS

All serious adverse experiences and adverse reactions observed in patients wearing these lenses or experienced with these lenses should be reported to:

Johnson & Johnson Vision Care, Inc. 7500 Centurion Parkway Jacksonville, FL 32256 USA Tel: 1-800-843-2020 www.acutue.com

27

CR-5945, V9.0




Johnson & Johnson Vision Care, Inc. 7500 Centurion Parkway Jacksonville, FL 32256 USA Tel: 1-800-843-2020 www.acuvue.com



©Johnson & Johnson Vision Care, Inc. 2017 In Canada: Johnson & Johnson Vision Care division of Johnson & Johnson Inc. In USA: Johnson & Johnson Vision Care, Inc. Printed In USA Revision date: 07/17 Revision number: M-07-17-02

1-DAY ACUVUE® MOIST and LACREON® are Trademarks of Johnson & Johnson Vision Care, Inc.

CR-5945, V9.0


## APPENDIX D: PRESBYOPIC SYMPTOMS QUESTIONNAIRE



## APPENDIX E: OCULAR DOMINANCE



## APPENDIX F: TEST LENS FITTING GUIDE





# APPENDIX G: NON-INVASIVE TEAR BREAK-UP TIME (NITBUT) NON-INVASIVE TEAR BREAK-UP TIME



## APPENDIX H: LOGMAR VISUAL ACUITY



## APPENDIX I: RANDOT STEREOPSIS



## APPENDIX J: UNILATERAL COVER TEST



## APPENDIX K: FIXATION DISPARITY



# APPENDIX L: DISTANCE CONTRAST THRESHOLD DISTANCE CONTRAST THRESHOLD



## APPENDIX M: BLUR TOLERANCE TESTING





## APPENDIX N: PERSONALITY TEST (BIG 5)



## APPENDIX O: PRE-FIT INTERVIEW



## **APPENDIX P: POST-FIT INTERVIEW**



## APPENDIX Q: MEASUREMENT OF LENS CENTRATION WITH MEDMONT TOPOGRAPHER






## APPENDIX R:

- DETERMINATION OF NEAR ADD
- LENS FITTING CHARACTERISTICS
- SUBJECT REPORTED OCULAR SYMPTOMS
- DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS
- BIOMICROSCOPY SCALE
- KERATOMETRY PROCEDURE
- MEASUREMENT OF COAS WAVEFRONT ABBERATIONS
- LENS INSERTION AND REMOVAL
- WAM-5500 ON-AXIS AUTO REFRACTION MEASUREMENT

## DETERMINATION OF NEAR ADD



















#### LENS FITTING CHARACTERISTICS











CR-5945, V9.0





#### SUBJECT REPORTED OCULAR SYMPTOMS



# DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS


















### BIOMICROSCOPY SCALE









CR-5945, V9.0








#### KERATOMETRY PROCEDURE



### MEASUREMENT OF COAS WAVEFRONT ABBERATIONS



CR-5945, V9.0








CR-5945, V9.0












### LENS INSERTION AND REMOVAL

Title: Lens Insertion and Removal

Document Type: Work Instructions

Document Number: Revision Number: 2





| Title: | WAM-5500 On-axis Auto Refraction Measurement | |
|---|---|---|
| Document Type: | <b>Clinical Test Procedure</b> | 75 |
| <b>Document Number:</b> | | Revision Number: 3 |
| | - | |
| | · | |


# MEASURING PUPIL DIAMETER WITH NEUROPTICS VIP-300 VARIABLE PUPILLOMETER










#### PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE

Protocol Number and Title: CR-5945, Characterizing Successful Myopic Multifocal Contact Lens Wearers

Version and Date: 9.0 Amendment 8, 20 December 2019

I have read and understand the protocol specified above and agree on its content.

I agree to conduct this study according to ISO 14155,<sup>1</sup> GCP and ICH guidelines,<sup>2</sup> the Declaration of Helsinki,<sup>3</sup> United States (US) Code of Federal Regulations (CFR),<sup>4</sup> and the pertinent individual country laws/regulations and to comply with its obligations, participant to ethical and safety considerations. The Principal Investigator is responsible for ensuring that all clinical site personnel, including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

I will assure that no deviation from, or changes to the protocol will take place without prior agreement from the Sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial Subjects.

I am responsible for ensuring that all clinical site personnel including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

All clinical site personnel involved in the conduct of this study have completed Human Subjects Protection Training.

I agree to ensure that all clinical site personnel involved in the conduct of this study are informed about their obligations in meeting the above commitments.

I shall not disclose the information contained in this protocol or any results obtained from this study without written authorization.

| Principal Investigator: | | |
|-------------------------|------------------------------------------|------|
| - | Signature | Date |
| | N 1 | |
| | Name and Professional Position (Printed) | |
| Institution/Site: | | |
| | Institution/Site Name | |
| | Institution/Site Address | |